CLINICAL TRIAL: NCT02747927
Title: Phase III, Double-Blind, Randomized, Placebo-Controlled Trial to Investigate the Efficacy, Safety and Immunogenicity of a Tetravalent Dengue Vaccine (TDV) Administered Subcutaneously in Healthy Children Aged 4 - 16 Years Old
Brief Title: Efficacy, Safety and Immunogenicity of Takeda's Tetravalent Dengue Vaccine (TDV) in Healthy Children
Acronym: TIDES
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DEN-301; U1111-1166-8401 (Registry Identifier: WHO); PHRR150522-001010 (Registry Identifier: PHRR); 2018-003979-34 (Registry Identifier: EudraCT)
Record Dates: First submitted 2016-04-14; First posted 2016-04-22 (Estimated); Results first posted 2021-08-18 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Healthy Volunteers
Keywords: Drug therapy
MeSH Terms: interventions — Dengue Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Participants received placebo-matching TDV, 0.5 milliliters (mL), subcutaneous (SC) injection on Day 1 (Month 0) and Day 90 (Month 3) in Part 1 of the study. Participants eligible for Booster Phase received placebo matching TDV, SC injection on Day 1 booster [b] (Month 0b) in Part 4 of the study based on the randomization code applied in Part 1 of the study.
  Interventions: Drug: Placebo
- Tetravalent Dengue Vaccine (TDV) 0.5 mL (Experimental): Participants received TDV, 0.5 mL, SC injection on Day 1 (Month 0) and Day 90 (Month 3) in Part 1 of the study. Participants eligible for Booster Phase received TDV, SC injection on Day 1b (Month 0b) in Part 4 of the study based on the randomization code applied in Part 1 of the study.
  Interventions: Biological: Tetravalent Dengue Vaccine (TDV)

INTERVENTIONS:
Drug: Placebo — TDV placebo-matching SC injection.
  Arms: Placebo
Biological: Tetravalent Dengue Vaccine (TDV) — TDV SC injection.
  Arms: Tetravalent Dengue Vaccine (TDV) 0.5 mL

SUMMARY:
The main purpose of this study is to evaluate the efficacy of 2 doses of Tetravalent Dengue Vaccine Candidate (TDV) in preventing symptomatic dengue fever of any severity and due to any of the four dengue virus serotypes in 4 to 16 year old participants.

DETAILED DESCRIPTION:
The vaccine being tested in this study is Takeda's Tetravalent Dengue Vaccine Candidate (TDV). TDV is being tested to protect people against dengue fever and to look at long-term safety results. This study will look at the success rate of TDV in preventing dengue fever (vaccine efficacy) and long-term side effects of the vaccine.

The study will be conducted in 5 parts. Part 1 will evaluate vaccine efficacy (VE) and will last a minimum of 15 months. Part 2 will be for an additional 6 months to evaluate VE. Part 3 will evaluate long-term safety by following participants for side effects and will last an additional 3 years. Part 4 will evaluate safety for 13 months post-booster vaccination. Part 5 will be the long-term safety follow-up for 1 year after completion of Part 4. Participants may be enrolled into a dry-run to commence and test febrile surveillance methodology; this dry-run part may be up to 10 months prior to receiving study injection, however, will not be applicable to all trials sites or participants.

Approximately 20,100 participants will be enrolled into the study and randomly assigned (by chance) to one of the two treatment groups-which will remain undisclosed to the participants and study doctors during the study (unless there is an urgent medical need):

* TDV 0.5 mL subcutaneous injection
* Placebo (dummy inactive subcutaneous injection) - this is a solution that looks like the study drug but has no active ingredient

All participants will receive a single injection of TDV or placebo on Day 1, Day 90. Participation in a booster phase will be offered to approximately 10,500 participants to receive (TDV or placebo) on Day 1b (Day 1 in booster phase). A subset of participants will be asked to record any local symptoms at the injection site (Pain, Erythema and Swelling) in a diary card for 7 days after each injection. The same subset of participants will also be asked to record any systemic symptoms (child <6 years: fever, irritability/fussiness, drowsiness, loss of appetite and child ≥6 years: fever, headache, asthenia, malaise and myalgia) in a diary card for 14 days after each injection.

This multi-center trial will be conducted worldwide. The overall time to participate in this study is approximately 7 years excluding the dry-run. Participants will make multiple visits to the clinic and will be contacted at least every week for the entire study duration.

ELIGIBILITY:
Inclusion Criteria:

1. Is aged 4 to 16 years, inclusive, at the time of randomization.
2. Is in good health at the time of entry into the trial as determined by medical history, physical examination (including vital signs) and clinical judgment of the Investigator.
3. The participant and/or the participant's parent/guardian signs and dates an assent/written informed consent form where applicable, and any required privacy authorization prior to the initiation of any trial procedures, after the nature of the trial has been explained according to local regulatory requirements.
4. Can comply with trial procedures and are available for the duration of follow-up.

Inclusion criteria for Booster Phase:

1. Is included in the per-protocol set (PPS) of the trial.
2. Was aged 4 to 11 years at the time of randomization in the study (Day 1 [Month 0]).

Exclusion Criteria:

1. Has febrile illness (temperature ≥38°C) or moderate or severe acute illness or infection at the time of randomization.
2. Has history of or any illness that, in the opinion of the Investigator, might interfere with the results of the trial or pose an additional risk to the participant due to participation in the trial.
3. Has received any other vaccine within 14 days (for inactivated vaccines) or 28 days (for live vaccines) prior to Day 1 (Month 0) or planning to receive any vaccine within 28 days after Day 1 (Month 0).
4. Has participated in any clinical trial with another investigational product 30 days prior to Day 1 (Month 0) or intent to participate in another clinical trial at any time during the conduct of this trial.
5. Has previously participated in any clinical trial of a dengue candidate vaccine, or previous receipt of a dengue vaccine.
6. Is first degree relative of individuals involved in trial conduct.
7. Females of childbearing potential who are sexually active, and who have not used any of the acceptable contraceptive methods for at least 2 months prior to Day 1 (Month 0).
8. Females of childbearing potential who are sexually active, and who refuse to use an acceptable contraceptive method up to 6 weeks post-second vaccination.
9. Deprived of freedom by administrative or court order, or in an emergency setting, or hospitalized involuntarily.
10. Current alcohol abuse or drug addiction that may interfere with the participant's ability to comply with trial procedures.
11. Identified as an employee of the Investigator or trial center, with direct involvement in the proposed trial or other trials under the direction of that Investigator or trial center.

Exclusion criteria for Booster Phase:

1. Receipt of any other vaccine within 14 days (for inactivated vaccines) or 28 days (for live vaccines) prior to Day 1b (Month 0b), or planning to receive any vaccine within 28 days after Day 1b (Month 0b).
2. Participation in any clinical trial with another investigational product at any time during participation in this trial or intent to participate in another clinical trial at any time during the conduct of the booster phase of this trial.

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20099 (Actual)
Dates: Start 2016-04-26 (Actual); Primary Completion 2018-07-11 (Actual); Study Completion 2024-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (28):
- Brazil (4):
  - Universidade Federal Do Espirito Santo Hospital Universitario Cassiano Antonio de Moraes HUCAM, Vitória, Espírito Santo
  - Associacao Obras Sociais Irma Dulce Hospital Santo Antonio, Salvador, Estado de Bahia
  - Universidade Federal de Mato Grosso do Sul, Campo Grande, Mato Grosso do Sul
  - Centro de Estudos e Pesquisa em Molestias Infecciosas LTDA (CPCLIN), Cidade Alta, Natal - RN
- Colombia (4):
  - Centro de Atencion e Investigacion Medica S.A - CAIMED - Aguazul - PPDS-PV, Aguazul, Casanare Department
  - Centro de Atencion e Investigacion Medica S.A - CAIMED - Yopal - PPDS-PV, Yopal, Casanare Department
  - Centro de Atencion e Investigacion Medica S.A. - CAIMED - Acacias - PPDS-PV, Acacías, Meta Department
  - Centro de Estudios em Infectologia Pediatrica SAS (CEIP S.A.S), Cali, San Fernando
- Dominican Republic (2):
  - Hospital Maternidad Nuestra Senora de Altagracia, Santo Domingo, Distrito Nacional Santo Domingo
  - Calle Alexander Fleming No. 90 Esquina 37, Ensanche La Fe, Santo Domingo, Distrito Nacional Santo Domingo
- Universidad Nacional Autonoma de Nicaragua, León, Nicaragua
- Panama (4):
  - Centro De Vacunacion Internacional, S.A. (Cevaxin), Panama City
  - Centro De Vacunacion Internacional, S.A. (Cevaxin) Sede 24 de Diciembre, Panama City
  - Centro De Vacunacion Internacional, S.A. (Cevaxin) Sede Plaza Carolina, Panama City
  - Centro De Vacunacion Internacional, S.A.(Cevaxin) - La Chorrera, Panama City
- Philippines (6):
  - Dela Salle Health Sciences Institute, Dasmariñas, Cavite
  - Philippines-AFRIMS Virology Research Unit, Cebu City, Cebu
  - Research Institute for Tropical Medicine, City of Muntinlupa
  - University of the Philippine Manila, Ermita
  - Las Pinas Health Center A, Las Piñas
  - Las Pinas Health Center D, Las Piñas
- Sri Lanka (4):
  - Lady Ridgeway Hospital for Children, Colombo
  - Colombo South Teaching Hospital, Dehiwala
  - Negombo General Hospital, Negombo
  - Colombo North Teaching Hospital, Ragama
- Thailand (3):
  - The Hospital for Tropical Diseases, Bangkok, Bangkok
  - Phramongkutklao Hospital, Bangkok, Bangkok
  - Srinagarind Hospital, Khon Kaen

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Rauscher M, Youard Z, Faccin A, Patel SS, Pang H, Zent O. Pregnancy outcomes following unintentional exposure to TAK-003, a live-attenuated tetravalent dengue vaccine. Expert Rev Vaccines. 2025 Dec;24(1):221-229. doi: 10.1080/14760584.2025.2480297. Epub 2025 Mar 27. PMID 40099800
- [Derived] Borja-Tabora C, Fernando L, Lopez Medina E, Reynales H, Rivera L, Saez-Llorens X, Sirivichayakul C, Yu D, Folschweiller N, Moss KJ, Rauscher M, Tricou V, Zhao Y, Biswal S. Immunogenicity, Safety, and Efficacy of a Tetravalent Dengue Vaccine in Children and Adolescents: An Analysis by Age Group. Clin Infect Dis. 2025 Feb 5;80(1):199-206. doi: 10.1093/cid/ciae369. PMID 38995684
- [Derived] Sirivichayakul C, Biswal S, Saez-Llorens X, Lopez-Medina E, Borja-Tabora C, Bravo L, Kosalaraksa P, Alera MT, Reynales H, Rivera L, Watanaveeradej V, Yu D, Espinoza F, Dietze R, Fernando L, Wickramasinghe VP, Moreira ED Jr, Fernando AD, Gunasekera D, Luz K, Venancio da Cunha R, Oliveira AL, Rauscher M, Fan H, Borkowski A, Escudero I, Tuboi S, Lloyd E, Tricou V, Folschweiller N, LeFevre I, Vargas LM, Wallace D; TIDES Study Group. Efficacy and Safety of a Tetravalent Dengue Vaccine (TAK-003) in Children With Prior Japanese Encephalitis or Yellow Fever Vaccination. J Infect Dis. 2024 Dec 16;230(6):e1214-e1225. doi: 10.1093/infdis/jiae222. PMID 38682569
- [Derived] Tricou V, Yu D, Reynales H, Biswal S, Saez-Llorens X, Sirivichayakul C, Lopez P, Borja-Tabora C, Bravo L, Kosalaraksa P, Vargas LM, Alera MT, Rivera L, Watanaveeradej V, Dietze R, Fernando L, Wickramasinghe VP, Moreira ED Jr, Fernando AD, Gunasekera D, Luz K, Oliveira AL, Tuboi S, Escudero I, Hutagalung Y, Lloyd E, Rauscher M, Zent O, Folschweiller N, LeFevre I, Espinoza F, Wallace D. Long-term efficacy and safety of a tetravalent dengue vaccine (TAK-003): 4.5-year results from a phase 3, randomised, double-blind, placebo-controlled trial. Lancet Glob Health. 2024 Feb;12(2):e257-e270. doi: 10.1016/S2214-109X(23)00522-3. PMID 38245116
- [Derived] Saez-Llorens X, Biswal S, Borja-Tabora C, Fernando L, Liu M, Wallace D, Folschweiller N, Reynales H, LeFevre I; TIDES Study Group. Effect of the Tetravalent Dengue Vaccine TAK-003 on Sequential Episodes of Symptomatic Dengue. Am J Trop Med Hyg. 2023 Mar 6;108(4):722-726. doi: 10.4269/ajtmh.22-0673. Print 2023 Apr 5. PMID 36878213
- [Derived] Rivera L, Biswal S, Saez-Llorens X, Reynales H, Lopez-Medina E, Borja-Tabora C, Bravo L, Sirivichayakul C, Kosalaraksa P, Martinez Vargas L, Yu D, Watanaveeradej V, Espinoza F, Dietze R, Fernando L, Wickramasinghe P, Duarte MoreiraJr E, Fernando AD, Gunasekera D, Luz K, Venancioda Cunha R, Rauscher M, Zent O, Liu M, Hoffman E, LeFevre I, Tricou V, Wallace D, Alera M, Borkowski A. Three-year Efficacy and Safety of Takeda's Dengue Vaccine Candidate (TAK-003). Clin Infect Dis. 2022 Aug 24;75(1):107-117. doi: 10.1093/cid/ciab864. PMID 34606595
- [Derived] Biswal S, Borja-Tabora C, Martinez Vargas L, Velasquez H, Theresa Alera M, Sierra V, Johana Rodriguez-Arenales E, Yu D, Wickramasinghe VP, Duarte Moreira E Jr, Fernando AD, Gunasekera D, Kosalaraksa P, Espinoza F, Lopez-Medina E, Bravo L, Tuboi S, Hutagalung Y, Garbes P, Escudero I, Rauscher M, Bizjajeva S, LeFevre I, Borkowski A, Saez-Llorens X, Wallace D; TIDES study group. Efficacy of a tetravalent dengue vaccine in healthy children aged 4-16 years: a randomised, placebo-controlled, phase 3 trial. Lancet. 2020 May 2;395(10234):1423-1433. doi: 10.1016/S0140-6736(20)30414-1. Epub 2020 Mar 17. PMID 32197105
- [Derived] Biswal S, Reynales H, Saez-Llorens X, Lopez P, Borja-Tabora C, Kosalaraksa P, Sirivichayakul C, Watanaveeradej V, Rivera L, Espinoza F, Fernando L, Dietze R, Luz K, Venancio da Cunha R, Jimeno J, Lopez-Medina E, Borkowski A, Brose M, Rauscher M, LeFevre I, Bizjajeva S, Bravo L, Wallace D; TIDES Study Group. Efficacy of a Tetravalent Dengue Vaccine in Healthy Children and Adolescents. N Engl J Med. 2019 Nov 21;381(21):2009-2019. doi: 10.1056/NEJMoa1903869. Epub 2019 Nov 6. PMID 31693803
- See also: To obtain more information about this study, click this link. — https://clinicaltrials.takeda.com/study-detail/5f6b60224db2bf003ab49693?idFilter=%5B%22DEN-301%22%5D

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at various investigative sites globally from 26 April 2016 to 28 June 2024.
Pre-assignment Details: Healthy children and adolescents were randomized in a 2:1 ratio to receive either tetravalent dengue vaccine (TDV) or placebo followed by a booster vaccination.
Groups:
- Placebo: Participants received placebo-matching TDV, 0.5 milliliter (mL), subcutaneous (SC) injection on Day 1 (Month 0) and Day 90 (Month 3) in Part 1 of the study. Participants eligible for Booster Phase received placebo matching TDV, SC injection on Day 1b (Month 0b) in Part 4 of the study based on the randomization code applied in Part 1 of the study.
- TDV 0.5 mL: Participants received TDV, 0.5 mL, SC injection on Day 1 (Month 0) and Day 90 (Month 3) in Part 1 of the study. Participants eligible for Booster Phase received TDV, SC injection on Day 1b (Month 0b) in Part 4 of the study based on the randomization code applied in Part 1 of the study.
Period: Part 1: Vaccine Efficacy (Months 0-15)
Arm/Group | Placebo | TDV 0.5 mL
Started | 6698 | 13401
Safety Set (Safety Set included all randomized participants who received at least 1 dose of the trial vaccines (TDV or placebo).) | 6687 | 13380
Treatment Misallocations (These are participants who received the wrong study vaccination, i.e. instead of Placebo/Placebo or TDV/TDV for first and second vaccination, they received a mix of TDV and Placebo. These participants are not included in the Placebo or TDV arm of the Safety Set and were separately analyzed for selected summary tables only.) | 1 | 3
Completed (Number of participants who had not discontinued from the trial at the end of Part 1.) | 6520 | 13035
Not Completed | 178 | 366
Not completed — Adverse Event | 5 | 14
Not completed — Lost to Follow-up | 13 | 26
Not completed — Pregnancy | 19 | 42
Not completed — Protocol Violation | 2 | 5
Not completed — Withdrawal by Participant and/or Participants Parent/Guardian | 131 | 260
Not completed — Without Adult Consent in Place | 1 | 4
Not completed — Reason not Specified | 7 | 15
Period: Part 2: Additional VE (Months 16-21)
Arm/Group | Placebo | TDV 0.5 mL
Started | 6520 | 13035
Completed (Number of participants who had not discontinued from the trial at the end of Part 2.) | 6488 | 12963
Not Completed | 32 | 72
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 4 | 8
Not completed — Pregnancy | 11 | 17
Not completed — Withdrawal by Participant&/ortheir Parent/Guardian | 13 | 33
Not completed — Without Adult Consent in Place | 1 | 7
Not completed — Reason Not Specified | 3 | 6
Period: Part 3: Long Term Safety & VE (3 Years)
Arm/Group | Placebo | TDV 0.5 mL
Started | 6488 | 12963
Completed (Number of participants who had not discontinued from the trial at the end of Part 3.) | 6080 | 12179
Not Completed | 408 | 784
Not completed — Adverse Event | 6 | 10
Not completed — Lost to Follow-up | 67 | 149
Not completed — Pregnancy | 120 | 228
Not completed — Protocol Violation | 1 | 2
Not completed — Withdrawal by Participant and/or Participants Parent/Guardian | 119 | 227
Not completed — Without Adult Consent in Place | 82 | 150
Not completed — Reason Not Specified | 13 | 18
Period: Part 4: Booster VE & Safety (13 Months)
Arm/Group | Placebo | TDV 0.5 mL
Started (Only participants from the PPS who were 4 to 11 years of age at the time of randomization in the trial on Day 1 (Month 0) can participate in the booster phase of this trial.) | 2986 | 5991
Safety Set - Booster (Safety Set - Booster (SS-B) included all participants who received the booster dose of the trial vaccine (TDV or placebo).) | 2985 | 5990
Treatment-Misallocations (These are participants who received the wrong study vaccination during the booster. These participants are not included in the Placebo or the TDV arm of the Safety Set and were separately analyzed for selected summary tables only.) | 1 | 1
Completed (Number of participants who had not discontinued from the trial at the end of Part 4.) | 2940 | 5890
Not Completed | 46 | 101
Not completed — Adverse Event | 1 | 3
Not completed — Lost to Follow-up | 4 | 13
Not completed — Pregnancy | 8 | 15
Not completed — Withdrawal by Participant and/or Participants Parent/Guardian | 29 | 60
Not completed — Without Adult Consent in Place | 0 | 1
Not completed — Reason Not Specified | 4 | 9
Period: Part 5: Booster VE & Safety (1 Year)
Arm/Group | Placebo | TDV 0.5 mL
Started | 2940 | 5890
Completed | 2842 | 5672
Not Completed | 98 | 218
Not completed — Adverse Event | 0 | 3
Not completed — Lost to Follow-up | 8 | 30
Not completed — Pregnancy | 18 | 27
Not completed — Withdrawal by Subject | 18 | 40
Not completed — Without Adult Consent in Place | 14 | 29
Not completed — Reason Not Specified | 40 | 89

BASELINE CHARACTERISTICS:
Population: Per-Protocol Set (PPS) included all participants in the Full Analysis Set (FAS) who had no major protocol violations. FAS included all randomized participants who received at least 1 dose of the trial vaccines.
Groups:
- Placebo: Participants received placebo-matching TDV, 0.5 mL, SC injection on Day 1 (Month 0) and Day 90 (Month 3) in Part 1 of the study. Participants eligible for Booster Phase received placebo matching TDV, SC injection on Day 1b (Month 0b) in Part 4 of the study based on the randomization code applied in Part 1 of the study.
- Total: Total of all reporting groups
Arm/Group | Placebo | TDV 0.5 mL | Total
Number analyzed (Participants) | 6317 | 12704 | 19021
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.6 (3.34) | 9.6 (3.35) | 9.6 (3.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3098 | 6314 | 9412
  Male | 3219 | 6390 | 9609
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2379 | 4821 | 7200
  Asian | 2934 | 5888 | 8822
  Black or African American | 708 | 1353 | 2061
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
  White | 131 | 284 | 415
  More than one race or Unknown | 164 | 356 | 520
Region of Enrollment [Count of Participants; unit: Participants]
  Brazil | 504 | 1091 | 1595
  Colombia | 1155 | 2268 | 3423
  Dominican Republic | 533 | 1007 | 1540
  Nicaragua | 239 | 512 | 751
  Panama | 944 | 1930 | 2874
  Philippines | 1306 | 2554 | 3860
  Sri Lanka | 683 | 1368 | 2051
  Thailand | 953 | 1974 | 2927
Height [Mean (Standard Deviation); unit: cm] — Population: Number analyzed is number of participants with data available for height at Baseline.
  cm
    number analyzed (Participants) | 6313 | 12696 | 19009
    (all) | 134.87 (18.976) | 134.84 (19.151) | 134.85 (19.092)
Weight [Mean (Standard Deviation); unit: kg] — Population: Number analyzed is number of participants with data available for weight at Baseline.
  kg
    number analyzed (Participants) | 6317 | 12697 | 19014
    (all) | 33.77 (14.506) | 33.98 (14.951) | 33.91 (14.805)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI=weight (kg)/[height (m)^2]. Population: Number analyzed is number of participants with data available for BMI at Baseline.
  kg/m^2
    number analyzed (Participants) | 6313 | 12689 | 19002
    (all) | 17.67 (3.645) | 17.76 (3.831) | 17.73 (3.770)

OUTCOME MEASURES:

1. Primary Outcome: Vaccine Efficacy (VE) of Two Doses of Tetravalent Dengue Vaccine Candidate (TDV) in Preventing Virologically-Confirmed Dengue Fever Induced by Any Dengue Serotype
Description: The VE is defined as 1 - (λv/λc), where λv and λc denote the hazard rates for the TDV and placebo arms, respectively. A virologically-confirmed dengue case is defined as febrile illness (defined as temperature ≥38°C on any 2 of 3 consecutive days) or illness clinically suspected to be dengue by the Investigator with a positive serotype-specific reverse transcriptase polymerase chain reaction (RT-PCR). The primary endpoint of VE was assessed using the number of virologically-confirmed dengue fever cases that occurred during Part 1.
Time Frame: 30 days post-second vaccination (Day 120 [Month 4]) until the end of Part 1 (Month 15) when at least 120 cases of dengue fever were confirmed and minimum duration of participant follow-up was 12 months post-second vaccination
Population: PPS included all participants in the FAS who had no major protocol violations. FAS included all randomized participants who received at least 1 dose of the trial vaccines. Overall number of participants analyzed is the number of participants with data available for analyses.
Measure: Number; unit: number of cases
Arm/Group | Placebo | TDV 0.5 mL
Number analyzed (Participants) | 6316 | 12700
number of cases | 149 | 61
Statistical Analysis 1: Comparison: Placebo vs TDV 0.5 mL; Assuming true VE of 60% and, virologically confirmed cases of dengue fever induced by any dengue serotype occurring from 30 days post 2nd vaccination (Day 120) until end of Part 1 would provide at least 90% power to rule out vaccine effect of ≤25%; Test type: Other; p < 0.001, Cox Proportional Hazard Model — Statistical significance was concluded if the lower bound of the 95% CI for the VE was above 25%. Since the hypotheses was tested in a confirmatory manner at a 2-sided significance level of 5%, the calculated p-value was compared with 0.025; VE = 80.2, 95% CI 2-sided [73.3 to 85.3] — VE and 95% CIs was estimated from Cox proportional hazard model with investigational product as a factor, adjusted for age, and stratified by region

2. Secondary Outcome: VE of Two Doses of TDV in Preventing Hospitalization Due to Virologically-Confirmed Dengue Fever Induced by Any Dengue Serotype
Description: VE is defined as 1 - (λv/λc), where λv and λc denote the hazard rates for the TDV and placebo arms, respectively. A virologically-confirmed dengue case is defined as febrile illness (defined as temperature ≥38°C on any 2 of 3 consecutive days) or illness clinically suspected to be dengue by the Investigator with a positive serotype-specific RT-PCR. VE was assessed using the number of cases requiring hospitalization due to virologically-confirmed dengue fever that occurred during Part 1 and Part 2.
Time Frame: From 30 days post-second vaccination (Day 120 [Month 4]) until the end of Part 2 (Month 21)
Population: as for outcome 1
Measure: Number; unit: number of cases
Arm/Group | Placebo | TDV 0.5 mL
Number analyzed (Participants) | 6316 | 12700
number of cases | 66 | 13
Statistical Analysis 1: Comparison: Placebo vs TDV 0.5 mL; Test type: Other; p < 0.001, Cox Proportional Hazard Model — Statistical significance was concluded if the lower bound of the 95% CI for the VE was above 0%. Since the hypotheses was tested in a confirmatory manner at a 2-sided significance level of 5%, the calculated p-value was compared with 0.025; VE = 90.4, 95% CI 2-sided [82.6 to 94.7] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: VE of Two Doses of TDV in Preventing Virologically-Confirmed Dengue Fever Induced by Each Dengue Serotype
Description: VE is defined as 1 - (λv/λc), where λv and λc denote the hazard rates for the TDV and placebo arms, respectively. A virologically-confirmed dengue case is defined as febrile illness (defined as temperature ≥38°C on any 2 of 3 consecutive days) or illness clinically suspected to be dengue by the Investigator with a positive serotype-specific RT-PCR. VE was assessed using the number of virologically-confirmed dengue fever cases that occurred during Part 1 and Part 2.
Time Frame: From 30 days post-second vaccination (Day 120 [Month 4]) until the end of Part 2 (Month 21)
Population: as for outcome 1
Measure: Number; unit: number of cases
Arm/Group | Placebo | TDV 0.5 mL
Number analyzed (Participants) | 6316 | 12700
number of cases
  DENV-1 | 62 | 38
  DENV-2 | 80 | 8
  DENV-3 | 60 | 63
  DENV-4 | 5 | 5
Statistical Analysis 1: Comparison: Placebo vs TDV 0.5 mL; DENV-1; Test type: Other; Cox Proportional Hazard Model; VE = 69.8, 95% CI 2-sided [54.8 to 79.9] — VE and two-sided 95% CIs are estimated from a Cox proportional hazard model with investigational product as a factor, adjusted for age, and stratified by region
Statistical Analysis 2: Comparison: Placebo vs TDV 0.5 mL; DENV-2; Test type: Other; Cox Proportional Hazard Model; VE = 95.1, 95% CI 2-sided [89.9 to 97.6] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs TDV 0.5 mL; DENV-3; Test type: Other; Cox Proportional Hazard Model; VE = 48.8, 95% CI 2-sided [27.1 to 64.1] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs TDV 0.5 mL; DENV-4; Test type: Other; Cox Proportional Hazard Model; VE = 50.9, 95% CI 2-sided [-69.7 to 85.8] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: VE of Two Doses of TDV in Preventing Virologically-Confirmed Dengue Fever Induced by Any Dengue Serotype in Participants Dengue Seronegative at Baseline
Description: as for outcome 3
Time Frame: From 30 days post-second vaccination (Day 120 [Month 4]) until the end of Part 2 (Month 21)
Population: PPS included all participants in the FAS who had no major protocol violations. FAS included all randomized participants who received at least 1 dose of the trial vaccines. Overall number of participants analyzed is the number of participants with seronegative baseline status and with data available for analyses.
Measure: Number; unit: number of cases
Arm/Group | Placebo | TDV 0.5 mL
Number analyzed (Participants) | 1726 | 3531
number of cases | 56 | 39
Statistical Analysis 1: Comparison: Placebo vs TDV 0.5 mL; Test type: Other; Cox Proportional Hazard Model; VE = 66.2, 95% CI 2-sided [49.1 to 77.5] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: VE of Two Doses of TDV in Preventing Virologically-Confirmed Dengue Fever Induced by Any Dengue Serotype in Participants Dengue Seropositive at Baseline
Description: as for outcome 3
Time Frame: From 30 days post-second vaccination (Day 120 [Month 4]) until the end of Part 2 (Month 21)
Population: PPS included all participants in the FAS who had no major protocol violations. FAS included all randomized participants who received at least 1 dose of the trial vaccines. Overall number of participants analyzed is the number of participants with seropositive baseline status and with data available for analyses.
Measure: Number; unit: number of cases
Arm/Group | Placebo | TDV 0.5 mL
Number analyzed (Participants) | 4589 | 9167
number of cases | 150 | 75
Statistical Analysis 1: Comparison: Placebo vs TDV 0.5 mL; Test type: Other; Cox Proportional Hazard Model; VE = 76.1, 95% CI 2-sided [68.5 to 81.9] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: VE of Two Doses of TDV in Preventing Virologically-Confirmed Severe Dengue Fever Induced by Any Dengue Serotype
Description: VE is defined as 1 - (λv/λc), where λv and λc denote the hazard rates for the TDV and placebo arms, respectively. A virologically-confirmed dengue case is defined as febrile illness (defined as temperature ≥38°C on any 2 of 3 consecutive days) or illness clinically suspected to be dengue by the Investigator with a positive serotype-specific RT-PCR. Severe cases were determined by Adjudication Committee. VE was assessed using the number of severe cases due to virologically-confirmed dengue fever that occurred during Part 1 and Part 2.
Time Frame: From 30 days post-second vaccination (Day 120 [Month 4]) until the end of Part 2 (Month 21)
Population: as for outcome 1
Measure: Number; unit: number of cases
Arm/Group | Placebo | TDV 0.5 mL
Number analyzed (Participants) | 6316 | 12700
number of cases | 1 | 2
Statistical Analysis 1: Comparison: Placebo vs TDV 0.5 mL; Test type: Other; Cox Proportional Hazard Model; VE = 2.2, 95% CI 2-sided [-978.5 to 91.1] — [estimate comment as in outcome 3, analysis 1]

7. Secondary Outcome: Percentage of Participants With Solicited Local Injection Site Adverse Events (AEs) by Severity in the Safety Set Immunogenicity Subset
Description: Solicited local AEs at injection site are defined as pain, erythema and swelling that occurred within 7 days after each vaccination. The participant/legal guardian recorded the severity of each AE (except erythema and swelling) according to the diary card instruction as none, mild, moderate, or severe. Severity grades for erythema and swelling were derived from the recorded diameters. Percentages were rounded off to the nearest single decimal place except the data points where rounding-up may lead to data misinterpretation.
Time Frame: Days 1 through 7 after each vaccination
Population: The Safety Set (SS)- Immunogenicity Subset included all randomized participants in the safety/immunogenicity subset who received at least 1 dose of the trial vaccines (TDV or placebo). Number analyzed is the number of participants with data available for analyses for the specified category.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TDV 0.5 mL
Number analyzed (Participants) | 1329 | 2663
percentage of participants
  Children of Age <6 Years; After First Vaccination; Pain: Mild: number analyzed (Participants) | 169 | 327
  Children of Age <6 Years; After First Vaccination; Pain: Mild | 19.5 | 21.1
  Children of Age <6 Years; After First Vaccination; Pain: Moderate: number analyzed (Participants) | 169 | 327
  Children of Age <6 Years; After First Vaccination; Pain: Moderate | 1.2 | 2.1
  Children of Age <6 Years; After First Vaccination; Pain: Severe: number analyzed (Participants) | 169 | 327
  Children of Age <6 Years; After First Vaccination; Pain: Severe | 0.6 | 0.3
  Children of Age <6 Years; After First Vaccination; Erythema; Mild: number analyzed (Participants) | 169 | 324
  Children of Age <6 Years; After First Vaccination; Erythema; Mild | 0.6 | 0.6
  Children of Age <6 Years; After First Vaccination; Erythema; Moderate: number analyzed (Participants) | 169 | 324
  Children of Age <6 Years; After First Vaccination; Erythema; Moderate | 0 | 0.6
  Children of Age <6 Years; After First Vaccination; Erythema; Severe: number analyzed (Participants) | 169 | 324
  Children of Age <6 Years; After First Vaccination; Erythema; Severe | 0 | 0
  Children of Age <6 Years; After First Vaccination; Swelling; Mild: number analyzed (Participants) | 169 | 324
  Children of Age <6 Years; After First Vaccination; Swelling; Mild | 0.6 | 1.9
  Children of Age <6 Years; After First Vaccination; Swelling; Moderate: number analyzed (Participants) | 169 | 324
  Children of Age <6 Years; After First Vaccination; Swelling; Moderate | 0 | 0.9
  Children of Age <6 Years; After First Vaccination; Swelling; Severe: number analyzed (Participants) | 169 | 324
  Children of Age <6 Years; After First Vaccination; Swelling; Severe | 0 | 0
  Children of Age <6 Years; After Second Vaccination; Pain: Mild: number analyzed (Participants) | 165 | 324
  Children of Age <6 Years; After Second Vaccination; Pain: Mild | 13.3 | 18.2
  Children of Age <6 Years; After Second Vaccination; Pain: Moderate: number analyzed (Participants) | 165 | 324
  Children of Age <6 Years; After Second Vaccination; Pain: Moderate | 1.2 | 2.5
  Children of Age <6 Years; After Second Vaccination; Pain: Severe: number analyzed (Participants) | 165 | 324
  Children of Age <6 Years; After Second Vaccination; Pain: Severe | 0 | 0
  Children of Age <6 Years; After Second Vaccination; Erythema; Mild: number analyzed (Participants) | 165 | 322
  Children of Age <6 Years; After Second Vaccination; Erythema; Mild | 0 | 0.6
  Children of Age <6 Years; After Second Vaccination; Erythema; Moderate: number analyzed (Participants) | 165 | 322
  Children of Age <6 Years; After Second Vaccination; Erythema; Moderate | 0 | 0
  Children of Age <6 Years; After Second Vaccination; Erythema; Severe: number analyzed (Participants) | 165 | 322
  Children of Age <6 Years; After Second Vaccination; Erythema; Severe | 0 | 0
  Children of Age <6 Years; After Second Vaccination; Swelling; Mild: number analyzed (Participants) | 164 | 323
  Children of Age <6 Years; After Second Vaccination; Swelling; Mild | 0.6 | 0.9
  Children of Age <6 Years; After Second Vaccination; Swelling; Moderate: number analyzed (Participants) | 164 | 323
  Children of Age <6 Years; After Second Vaccination; Swelling; Moderate | 0 | 0.6
  Children of Age <6 Years; After Second Vaccination; Swelling; Severe: number analyzed (Participants) | 164 | 323
  Children of Age <6 Years; After Second Vaccination; Swelling; Severe | 0 | 0
  Children of Age >=6 Years; After First Vaccination; Pain: Mild: number analyzed (Participants) | 1143 | 2284
  Children of Age >=6 Years; After First Vaccination; Pain: Mild | 16.9 | 23.4
  Children of Age >=6 Years; After First Vaccination; Pain: Moderate: number analyzed (Participants) | 1143 | 2284
  Children of Age >=6 Years; After First Vaccination; Pain: Moderate | 2.2 | 3.9
  Children of Age >=6 Years; After First Vaccination; Pain: Severe: number analyzed (Participants) | 1143 | 2284
  Children of Age >=6 Years; After First Vaccination; Pain: Severe | 0.3 | 0.7
  Children of Age >=6 Years; After First Vaccination; Erythema; Mild: number analyzed (Participants) | 1140 | 2276
  Children of Age >=6 Years; After First Vaccination; Erythema; Mild | 0 | 1.0
  Children of Age >=6 Years; After First Vaccination; Erythema; Moderate: number analyzed (Participants) | 1140 | 2276
  Children of Age >=6 Years; After First Vaccination; Erythema; Moderate | 0 | 0
  Children of Age >=6 Years; After First Vaccination; Erythema; Severe: number analyzed (Participants) | 1140 | 2276
  Children of Age >=6 Years; After First Vaccination; Erythema; Severe | 0 | 0
  Children of Age >=6 Years; After First Vaccination; Swelling; Mild: number analyzed (Participants) | 1140 | 2272
  Children of Age >=6 Years; After First Vaccination; Swelling; Mild | 0.4 | 1.2
  Children of Age >=6 Years; After First Vaccination; Swelling; Moderate: number analyzed (Participants) | 1140 | 2272
  Children of Age >=6 Years; After First Vaccination; Swelling; Moderate | 0 | 0
  Children of Age >=6 Years; After First Vaccination; Swelling; Severe: number analyzed (Participants) | 1140 | 2272
  Children of Age >=6 Years; After First Vaccination; Swelling; Severe | 0 | 0
  Children of Age >=6 Years; After Second Vaccination Pain; Mild: number analyzed (Participants) | 1116 | 2251
  Children of Age >=6 Years; After Second Vaccination Pain; Mild | 10.7 | 19.7
  Children of Age >=6 Years; After Second Vaccination Pain; Moderate: number analyzed (Participants) | 1116 | 2251
  Children of Age >=6 Years; After Second Vaccination Pain; Moderate | 1.5 | 3.2
  Children of Age >=6 Years; After Second Vaccination Pain; Severe: number analyzed (Participants) | 1116 | 2251
  Children of Age >=6 Years; After Second Vaccination Pain; Severe | 0.3 | 0.6
  Children of Age >=6 Years; After Second Vaccination Erythema; Mild: number analyzed (Participants) | 1113 | 2248
  Children of Age >=6 Years; After Second Vaccination Erythema; Mild | 0.0898 | 0.9
  Children of Age >=6 Years; After Second Vaccination Erythema; Moderate: number analyzed (Participants) | 1113 | 2248
  Children of Age >=6 Years; After Second Vaccination Erythema; Moderate | 0 | 0
  Children of Age >=6 Years; After Second Vaccination Erythema; Severe: number analyzed (Participants) | 1113 | 2248
  Children of Age >=6 Years; After Second Vaccination Erythema; Severe | 0 | 0
  Children of Age >=6 Years; After Second Vaccination Swelling; Mild: number analyzed (Participants) | 1112 | 2246
  Children of Age >=6 Years; After Second Vaccination Swelling; Mild | 0.0899 | 0.6
  Children of Age >=6 Years; After Second Vaccination Swelling; Moderate: number analyzed (Participants) | 1112 | 2246
  Children of Age >=6 Years; After Second Vaccination Swelling; Moderate | 0 | 0
  Children of Age >=6 Years; After Second Vaccination Swelling; Severe: number analyzed (Participants) | 1112 | 2246
  Children of Age >=6 Years; After Second Vaccination Swelling; Severe | 0 | 0

8. Secondary Outcome: Percentage of Participants With Solicited Systemic Adverse Events (AEs) by Severity in the Safety Set Immunogenicity Subset
Description: Solicited systemic AEs in children (< 6 years) are defined as fever, irritability/fussiness, drowsiness and loss of appetite that occurred within 14 days after each vaccination. Solicited systemic AEs in children (≥ 6 years) are defined as fever, headache, asthenia, malaise and myalgia that occurred within 14 days after each vaccination. The participant/legal guardian recorded the severity of each AE (except fever) according to the diary card instruction as none, mild, moderate, or severe. Severity grades for fever were derived from the recorded body temperature measurements and presented using the proposed temperature increments published by the Brighton Collaboration. Percentages were rounded off to the nearest single decimal place except the data points where rounding-up may lead to data misinterpretation.
Time Frame: Days 1 through 14 after each vaccination on Day 1 (Month 0) and Day 90 (Month 3)
Population: The SS- Immunogenicity Subset included all randomized participants in the safety/immunogenicity subset who received at least 1 dose of the trial vaccines (TDV or placebo). Number analyzed is the number of participants with data available for analysis for the specified category.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TDV 0.5 mL
Number analyzed (Participants) | 1329 | 2663
percentage of participants
  Children of Age <6 Years; After First Vaccination; Irritability/Fussiness: Mild: number analyzed (Participants) | 169 | 325
  Children of Age <6 Years; After First Vaccination; Irritability/Fussiness: Mild | 8.3 | 7.7
  Children of Age <6 Years; After First Vaccination; Irritability/Fussiness: Moderate: number analyzed (Participants) | 169 | 325
  Children of Age <6 Years; After First Vaccination; Irritability/Fussiness: Moderate | 0.6 | 0.9
  Children of Age <6 Years; After First Vaccination; Irritability/Fussiness: Severe: number analyzed (Participants) | 169 | 325
  Children of Age <6 Years; After First Vaccination; Irritability/Fussiness: Severe | 0 | 0.3
  Children of Age <6 Years; After First Vaccination; Drowsiness; Mild: number analyzed (Participants) | 169 | 325
  Children of Age <6 Years; After First Vaccination; Drowsiness; Mild | 10.1 | 8.3
  Children of Age <6 Years; After First Vaccination; Drowsiness; Moderate: number analyzed (Participants) | 169 | 325
  Children of Age <6 Years; After First Vaccination; Drowsiness; Moderate | 0 | 2.2
  Children of Age <6 Years; After First Vaccination; Drowsiness; Severe: number analyzed (Participants) | 169 | 325
  Children of Age <6 Years; After First Vaccination; Drowsiness; Severe | 0 | 0.6
  Children of Age <6 Years; After First Vaccination; Loss of Appetite; Mild: number analyzed (Participants) | 169 | 325
  Children of Age <6 Years; After First Vaccination; Loss of Appetite; Mild | 7.1 | 12.3
  Children of Age <6 Years; After First Vaccination; Loss of Appetite; Moderate: number analyzed (Participants) | 169 | 325
  Children of Age <6 Years; After First Vaccination; Loss of Appetite; Moderate | 1.8 | 1.2
  Children of Age <6 Years; After First Vaccination; Loss of Appetite; Severe: number analyzed (Participants) | 169 | 325
  Children of Age <6 Years; After First Vaccination; Loss of Appetite; Severe | 0.6 | 0.6
  Children of Age <6 Years; After First Vaccination; Fever; 38.0-<38.5: number analyzed (Participants) | 153 | 311
  Children of Age <6 Years; After First Vaccination; Fever; 38.0-<38.5 | 3.3 | 3.9
  Children of Age <6 Years; After First Vaccination; Fever; 38.5-<39.0: number analyzed (Participants) | 153 | 311
  Children of Age <6 Years; After First Vaccination; Fever; 38.5-<39.0 | 2.0 | 1.9
  Children of Age <6 Years; After First Vaccination; Fever; 39.0-<39.5: number analyzed (Participants) | 153 | 311
  Children of Age <6 Years; After First Vaccination; Fever; 39.0-<39.5 | 2.0 | 1.9
  Children of Age <6 Years; After First Vaccination; Fever; 39.5-<40.0: number analyzed (Participants) | 153 | 311
  Children of Age <6 Years; After First Vaccination; Fever; 39.5-<40.0 | 0.7 | 1.0
  Children of Age <6 Years; After First Vaccination; Fever: >=40.0: number analyzed (Participants) | 153 | 311
  Children of Age <6 Years; After First Vaccination; Fever: >=40.0 | 0 | 0
  Children of Age <6 Years; After Second Vaccination; Irritability/Fussiness: Mild: number analyzed (Participants) | 143 | 284
  Children of Age <6 Years; After Second Vaccination; Irritability/Fussiness: Mild | 2.1 | 5.3
  Children of Age <6 Years; After Second Vaccination; Irritability/Fussiness: Moderate: number analyzed (Participants) | 143 | 284
  Children of Age <6 Years; After Second Vaccination; Irritability/Fussiness: Moderate | 0 | 0.4
  Children of Age <6 Years; After Second Vaccination; Irritability/Fussiness: Severe: number analyzed (Participants) | 143 | 284
  Children of Age <6 Years; After Second Vaccination; Irritability/Fussiness: Severe | 0 | 0.4
  Children of Age <6 Years; After Second Vaccination; Drowsiness; Mild: number analyzed (Participants) | 143 | 284
  Children of Age <6 Years; After Second Vaccination; Drowsiness; Mild | 4.9 | 6.0
  Children of Age <6 Years; After Second Vaccination; Drowsiness; Moderate: number analyzed (Participants) | 143 | 284
  Children of Age <6 Years; After Second Vaccination; Drowsiness; Moderate | 0 | 1.1
  Children of Age <6 Years; After Second Vaccination; Drowsiness; Severe: number analyzed (Participants) | 143 | 284
  Children of Age <6 Years; After Second Vaccination; Drowsiness; Severe | 0 | 0
  Children of Age <6 Years; After Second Vaccination; Loss of Appetite; Mild: number analyzed (Participants) | 143 | 284
  Children of Age <6 Years; After Second Vaccination; Loss of Appetite; Mild | 4.9 | 6.0
  Children of Age <6 Years; After Second Vaccination; Loss of Appetite; Moderate: number analyzed (Participants) | 143 | 284
  Children of Age <6 Years; After Second Vaccination; Loss of Appetite; Moderate | 0.7 | 1.1
  Children of Age <6 Years; After Second Vaccination; Loss of Appetite; Severe: number analyzed (Participants) | 143 | 284
  Children of Age <6 Years; After Second Vaccination; Loss of Appetite; Severe | 0.7 | 0.4
  Children of Age <6 Years; After Second Vaccination; Fever: 38.0-<38.5: number analyzed (Participants) | 158 | 313
  Children of Age <6 Years; After Second Vaccination; Fever: 38.0-<38.5 | 4.4 | 1.3
  Children of Age <6 Years; After Second Vaccination; Fever: 38.5-<39.0: number analyzed (Participants) | 158 | 313
  Children of Age <6 Years; After Second Vaccination; Fever: 38.5-<39.0 | 1.3 | 3.5
  Children of Age <6 Years; After Second Vaccination; Fever: 39.0-<39.5: number analyzed (Participants) | 158 | 313
  Children of Age <6 Years; After Second Vaccination; Fever: 39.0-<39.5 | 1.3 | 1.3
  Children of Age <6 Years; After Second Vaccination; Fever: 39.5-<40.0: number analyzed (Participants) | 158 | 313
  Children of Age <6 Years; After Second Vaccination; Fever: 39.5-<40.0 | 0 | 0.6
  Children of Age <6 Years; After Second Vaccination; Fever: 40.0-<40.5: number analyzed (Participants) | 158 | 313
  Children of Age <6 Years; After Second Vaccination; Fever: 40.0-<40.5 | 0.6 | 0.3
  Children of Age <6 Years; After Second Vaccination; Fever: >=40.5: number analyzed (Participants) | 158 | 313
  Children of Age <6 Years; After Second Vaccination; Fever: >=40.5 | 0 | 0
  Children of Age >=6 Years; After First Vaccination; Headache: Mild: number analyzed (Participants) | 1142 | 2284
  Children of Age >=6 Years; After First Vaccination; Headache: Mild | 17.8 | 17.5
  Children of Age >=6 Years; After First Vaccination; Headache: Moderate: number analyzed (Participants) | 1142 | 2284
  Children of Age >=6 Years; After First Vaccination; Headache: Moderate | 3.4 | 5.3
  Children of Age >=6 Years; After First Vaccination; Headache: Severe: number analyzed (Participants) | 1142 | 2284
  Children of Age >=6 Years; After First Vaccination; Headache: Severe | 1.7 | 1.8
  Children of Age >=6 Years; After First Vaccination; Asthenia: Mild: number analyzed (Participants) | 1142 | 2285
  Children of Age >=6 Years; After First Vaccination; Asthenia: Mild | 8.8 | 8.8
  Children of Age >=6 Years; After First Vaccination; Asthenia: Moderate: number analyzed (Participants) | 1142 | 2285
  Children of Age >=6 Years; After First Vaccination; Asthenia: Moderate | 2.8 | 2.8
  Children of Age >=6 Years; After First Vaccination; Asthenia: Severe: number analyzed (Participants) | 1142 | 2285
  Children of Age >=6 Years; After First Vaccination; Asthenia: Severe | 0.5 | 0.8
  Children of Age >=6 Years; After First Vaccination; Malaise: Mild: number analyzed (Participants) | 1142 | 2283
  Children of Age >=6 Years; After First Vaccination; Malaise: Mild | 11.1 | 11.8
  Children of Age >=6 Years; After First Vaccination; Malaise: Moderate: number analyzed (Participants) | 1142 | 2283
  Children of Age >=6 Years; After First Vaccination; Malaise: Moderate | 2.3 | 3.4
  Children of Age >=6 Years; After First Vaccination; Malaise: Severe: number analyzed (Participants) | 1142 | 2283
  Children of Age >=6 Years; After First Vaccination; Malaise: Severe | 0.8 | 1.0
  Children of Age >=6 Years; After First Vaccination; Muscle Pain: Mild: number analyzed (Participants) | 1142 | 2283
  Children of Age >=6 Years; After First Vaccination; Muscle Pain: Mild | 11.8 | 14.1
  Children of Age >=6 Years; After First Vaccination; Muscle Pain: Moderate: number analyzed (Participants) | 1142 | 2283
  Children of Age >=6 Years; After First Vaccination; Muscle Pain: Moderate | 1.9 | 2.9
  Children of Age >=6 Years; After First Vaccination; Muscle Pain: Severe: number analyzed (Participants) | 1142 | 2283
  Children of Age >=6 Years; After First Vaccination; Muscle Pain: Severe | 0.6 | 0.9
  Children of Age >=6 Years; After First Vaccination; Fever: 38.0-<38.5: number analyzed (Participants) | 1052 | 2088
  Children of Age >=6 Years; After First Vaccination; Fever: 38.0-<38.5 | 3.0 | 3.0
  Children of Age >=6 Years; After First Vaccination; Fever: 38.5-<39.0: number analyzed (Participants) | 1052 | 2088
  Children of Age >=6 Years; After First Vaccination; Fever: 38.5-<39.0 | 1.8 | 2.0
  Children of Age >=6 Years; After First Vaccination; Fever: 39.0-<39.5: number analyzed (Participants) | 1052 | 2088
  Children of Age >=6 Years; After First Vaccination; Fever: 39.0-<39.5 | 1.0 | 0.5
  Children of Age >=6 Years; After First Vaccination; Fever: 39.5-<40.0: number analyzed (Participants) | 1052 | 2088
  Children of Age >=6 Years; After First Vaccination; Fever: 39.5-<40.0 | 0.4 | 0.4
  Children of Age >=6 Years; After First Vaccination; Fever: 40.0-<40.5: number analyzed (Participants) | 1052 | 2088
  Children of Age >=6 Years; After First Vaccination; Fever: 40.0-<40.5 | 0.0951 | 0.0479
  Children of Age >=6 Years; After First Vaccination; Fever: 40.5-<41.0: number analyzed (Participants) | 1052 | 2088
  Children of Age >=6 Years; After First Vaccination; Fever: 40.5-<41.0 | 0.0951 | 0
  Children of Age >=6 Years; After First Vaccination; Fever: >=41.0: number analyzed (Participants) | 1052 | 2088
  Children of Age >=6 Years; After First Vaccination; Fever: >=41.0 | 0 | 0
  Children of Age >=6 Years; After Second Vaccination; Headache: Mild: number analyzed (Participants) | 1117 | 2248
  Children of Age >=6 Years; After Second Vaccination; Headache: Mild | 10.2 | 10.4
  Children of Age >=6 Years; After Second Vaccination; Headache: Moderate: number analyzed (Participants) | 1117 | 2248
  Children of Age >=6 Years; After Second Vaccination; Headache: Moderate | 2.9 | 3.5
  Children of Age >=6 Years; After Second Vaccination; Headache: Severe: number analyzed (Participants) | 1117 | 2248
  Children of Age >=6 Years; After Second Vaccination; Headache: Severe | 1.1 | 1.3
  Children of Age >=6 Years; After Second Vaccination; Asthenia: Mild: number analyzed (Participants) | 1117 | 2248
  Children of Age >=6 Years; After Second Vaccination; Asthenia: Mild | 5.6 | 6.6
  Children of Age >=6 Years; After Second Vaccination; Asthenia: Moderate: number analyzed (Participants) | 1117 | 2248
  Children of Age >=6 Years; After Second Vaccination; Asthenia: Moderate | 1.6 | 1.9
  Children of Age >=6 Years; After Second Vaccination; Asthenia: Severe: number analyzed (Participants) | 1117 | 2248
  Children of Age >=6 Years; After Second Vaccination; Asthenia: Severe | 0.4 | 0.7
  Children of Age >=6 Years; After Second Vaccination; Malaise: Mild: number analyzed (Participants) | 1117 | 2248
  Children of Age >=6 Years; After Second Vaccination; Malaise: Mild | 6.8 | 8.1
  Children of Age >=6 Years; After Second Vaccination; Malaise: Moderate: number analyzed (Participants) | 1117 | 2248
  Children of Age >=6 Years; After Second Vaccination; Malaise: Moderate | 1.8 | 1.9
  Children of Age >=6 Years; After Second Vaccination; Malaise: Severe: number analyzed (Participants) | 1117 | 2248
  Children of Age >=6 Years; After Second Vaccination; Malaise: Severe | 0.8 | 1.0
  Children of Age >=6 Years; After Second Vaccination; Muscle Pain: Mild: number analyzed (Participants) | 1117 | 2248
  Children of Age >=6 Years; After Second Vaccination; Muscle Pain: Mild | 7.6 | 10.7
  Children of Age >=6 Years; After Second Vaccination; Muscle Pain: Moderate: number analyzed (Participants) | 1117 | 2248
  Children of Age >=6 Years; After Second Vaccination; Muscle Pain: Moderate | 1.3 | 2.0
  Children of Age >=6 Years; After Second Vaccination; Muscle Pain: Severe: number analyzed (Participants) | 1117 | 2248
  Children of Age >=6 Years; After Second Vaccination; Muscle Pain: Severe | 0.4 | 0.9
  Children of Age >=6 Years; After Second Vaccination; Fever: 38.0-<38.5: number analyzed (Participants) | 1056 | 2142
  Children of Age >=6 Years; After Second Vaccination; Fever: 38.0-<38.5 | 3.4 | 2.0
  Children of Age >=6 Years; After Second Vaccination; Fever: 38.5-<39.0: number analyzed (Participants) | 1056 | 2142
  Children of Age >=6 Years; After Second Vaccination; Fever: 38.5-<39.0 | 1.2 | 1.5
  Children of Age >=6 Years; After Second Vaccination; Fever: 39.0-<39.5: number analyzed (Participants) | 1056 | 2142
  Children of Age >=6 Years; After Second Vaccination; Fever: 39.0-<39.5 | 1.1 | 0.7
  Children of Age >=6 Years; After Second Vaccination; Fever: 39.5-<40.0: number analyzed (Participants) | 1056 | 2142
  Children of Age >=6 Years; After Second Vaccination; Fever: 39.5-<40.0 | 0.4 | 0.5
  Children of Age >=6 Years; After Second Vaccination; Fever: 40.0-<40.5: number analyzed (Participants) | 1056 | 2142
  Children of Age >=6 Years; After Second Vaccination; Fever: 40.0-<40.5 | 0 | 0.0467
  Children of Age >=6 Years; After Second Vaccination; Fever: >=40.5: number analyzed (Participants) | 1056 | 2142
  Children of Age >=6 Years; After Second Vaccination; Fever: >=40.5 | 0 | 0

9. Secondary Outcome: Percentage of Participants With Any Unsolicited Adverse Events (AEs) in the Safety Set Immunogenicity Subset
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a trial vaccine; it does not necessarily have to have a causal relationship with trial vaccine administration. Unsolicited AEs are any AEs that are not solicited local or systemic AEs, as defined by this study. Percentages were rounded off to the nearest single decimal place.
Time Frame: Days 1 through 28 after each vaccination on Day 1 (Month 0) and Day 90 (Month 3)
Population: The SS-Immunogenicity Subset included all randomized participants in the safety/immunogenicity subset who received at least 1 dose of the trial vaccines (TDV or placebo). Number analyzed is the number of participants with data available for analysis for the specified category.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TDV 0.5 mL
Number analyzed (Participants) | 1329 | 2663
percentage of participants
  After First Vaccination | 11.6 | 11.1
  After Second Vaccination: number analyzed (Participants) | 1301 | 2606
  After Second Vaccination | 9.2 | 9.3

10. Secondary Outcome: Percentage of Participants With Serious Adverse Events (SAEs) During Parts 1 and 2
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a trial vaccine; it does not necessarily have to have a causal relationship with trial vaccine administration. A serious adverse event (SAE) is any untoward medical occurrence or effect that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability / incapacity, is a congenital anomaly / birth defect or is medically important due to other reasons than the above mentioned criteria. Percentages were rounded off to the nearest single decimal place. In the category 'Part 1 and 2 combined' participants are counted only once even if they experienced events in both Part 1 and Part 2 in order to yield total of unique participants who had SAEs.
Time Frame: From Day 1 until the end of Parts 1 (Month 15) and 2 (Month 21)
Population: The SS included all randomized participants who received at least one dose of the investigational product (IP) (TDV or placebo). Number analyzed is the number of participants at risk at the start of the specified analysis period.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TDV 0.5 mL
Number analyzed (Participants) | 6687 | 13380
percentage of participants
  Part 1 | 3.8 | 3.1
  Part 2: number analyzed (Participants) | 6519 | 13033
  Part 2 | 1.3 | 1.2
  Parts 1 and 2 Combined | 4.9 | 4.1

11. Secondary Outcome: Percentage of Participants With Fatal SAEs and SAEs Related to Study Drug During the First and Second Half of Part 3
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a trial vaccine; it does not necessarily have to have a causal relationship with trial vaccine administration. A SAE is any untoward medical occurrence or effect that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability / incapacity, is a congenital anomaly / birth defect or is medically important due to other reasons than the above mentioned criteria. Percentages were rounded off to the nearest single decimal place except the data points where rounding-up may lead to data misinterpretation.
Time Frame: First and Second half (18 months each) of Part 3 (up to 3 years, beginning at Month 22)
Population: The SS included all randomized participants who received at least one dose of the IP (TDV or placebo). Overall number of participants analyzed are the number of participants with data available for analyses. Number analyzed is the number of participants at risk at the start of the specified analysis period.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TDV 0.5 mL
Number analyzed (Participants) | 6487 | 12961
percentage of participants
  Fatal SAEs: First Half of Part 3 | 0.0308 | 0.0386
  SAEs Related to Study Drug: First Half of Part 3 | 0 | 0
  Fatal SAEs: Second Half of Part 3: number analyzed (Participants) | 6340 | 12660
  Fatal SAEs: Second Half of Part 3 | 0.0631 | 0.0474
  SAEs Related to Study Drug: Second Half of Part 3: number analyzed (Participants) | 6340 | 12660
  SAEs Related to Study Drug: Second Half of Part 3 | 0 | 0

12. Secondary Outcome: Seropositivity Rate for Each of the Four Dengue Serotypes in the Immunogenicity Subset
Description: Seropositivity rate, defined as the percentage of participants seropositive, is derived from the titers of dengue-neutralizing antibodies. Seropositivity is defined as a reciprocal neutralizing titer ≥10. The four DENV serotypes are DENV-1, DENV-2, DENV-3 and DENV-4. Percentages were rounded off to the nearest single decimal place except the data points where rounding-up may lead to data misinterpretation.
Time Frame: Pre-vaccination on Day 1 (Baseline), post-first vaccination on Month 1, pre-vaccination on Month 3; post-second vaccination at Months 4, 9 and 15, and then annually (up to 3 years)
Population: Per-Protocol Set for Immunogenicity (PPSI): all participants in Full Analysis Set for Immunogenicity (FASI) who had no major protocol violations. The FASI were based on FAS & included all randomized participants in subset for whom a valid pre-dosing and at least one valid post-dosing blood sample have been received for immunogenicity. Number analyzed is the number of participants with data available for analysis at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TDV 0.5 mL
Number analyzed (Participants) | 1247 | 2518
percentage of participants
  Baseline: DENV-1 | 65.5 | 64.3
  Baseline: DENV-2: number analyzed (Participants) | 1247 | 2517
  Baseline: DENV-2 | 70.3 | 69.6
  Baseline: DENV-3: number analyzed (Participants) | 1247 | 2517
  Baseline: DENV-3 | 63.7 | 63.5
  Baseline: DENV-4 | 63.2 | 63.5
  Month 1: DENV-1: number analyzed (Participants) | 1165 | 2353
  Month 1: DENV-1 | 65.0 | 98.0
  Month 1: DENV-2: number analyzed (Participants) | 1164 | 2353
  Month 1: DENV-2 | 70.0 | 99.5
  Month 1: DENV-3: number analyzed (Participants) | 1164 | 2353
  Month 1: DENV-3 | 64.0 | 98.7
  Month 1: DENV-4: number analyzed (Participants) | 1165 | 2353
  Month 1: DENV-4 | 62.7 | 97.1
  Month 3: DENV-1: number analyzed (Participants) | 1244 | 2515
  Month 3: DENV-1 | 66.9 | 97.1
  Month 3: DENV-2: number analyzed (Participants) | 1244 | 2515
  Month 3: DENV-2 | 71.2 | 99.7
  Month 3: DENV-3: number analyzed (Participants) | 1243 | 2515
  Month 3: DENV-3 | 63.6 | 98.1
  Month 3: DENV-4: number analyzed (Participants) | 1244 | 2515
  Month 3: DENV-4 | 63.6 | 97.3
  Month 4: DENV-1: number analyzed (Participants) | 1131 | 2262
  Month 4: DENV-1 | 67.6 | 99.8
  Month 4: DENV-2: number analyzed (Participants) | 1131 | 2262
  Month 4: DENV-2 | 71.8 | 99.912
  Month 4: DENV-3: number analyzed (Participants) | 1131 | 2262
  Month 4: DENV-3 | 65.0 | 99.9
  Month 4: DENV-4: number analyzed (Participants) | 1131 | 2262
  Month 4: DENV-4 | 65.2 | 99.912
  Month 9: DENV-1: number analyzed (Participants) | 1085 | 2196
  Month 9: DENV-1 | 67.5 | 98.3
  Month 9: DENV-2: number analyzed (Participants) | 1085 | 2196
  Month 9: DENV-2 | 73.5 | 100.0
  Month 9: DENV-3: number analyzed (Participants) | 1085 | 2196
  Month 9: DENV-3 | 65.2 | 98.8
  Month 9: DENV-4: number analyzed (Participants) | 1085 | 2196
  Month 9: DENV-4 | 65.2 | 99.0
  Month 15: DENV-1: number analyzed (Participants) | 1115 | 2213
  Month 15: DENV-1 | 67.7 | 97.6
  Month 15: DENV-2: number analyzed (Participants) | 1115 | 2214
  Month 15: DENV-2 | 70.4 | 99.955
  Month 15: DENV-3: number analyzed (Participants) | 1115 | 2215
  Month 15: DENV-3 | 64.3 | 97.7
  Month 15: DENV-4: number analyzed (Participants) | 1115 | 2215
  Month 15: DENV-4 | 66.0 | 98.4
  Year 1: DENV-1: number analyzed (Participants) | 942 | 1904
  Year 1: DENV-1 | 69.6 | 97.0
  Year 1: DENV-2: number analyzed (Participants) | 942 | 1904
  Year 1: DENV-2 | 72.0 | 99.9
  Year 1: DENV-3: number analyzed (Participants) | 942 | 1904
  Year 1: DENV-3 | 67.5 | 97.3
  Year 1: DENV-4: number analyzed (Participants) | 942 | 1904
  Year 1: DENV-4 | 68.6 | 98.3
  Year 2: DENV-1: number analyzed (Participants) | 955 | 1921
  Year 2: DENV-1 | 71.5 | 95.7
  Year 2: DENV-2: number analyzed (Participants) | 955 | 1921
  Year 2: DENV-2 | 73.7 | 99.948
  Year 2: DENV-3: number analyzed (Participants) | 955 | 1921
  Year 2: DENV-3 | 68.8 | 95.5
  Year 2: DENV-4: number analyzed (Participants) | 955 | 1921
  Year 2: DENV-4 | 70.7 | 98.0
  Year 3: DENV-1: number analyzed (Participants) | 1023 | 2049
  Year 3: DENV-1 | 72.5 | 94.9
  Year 3: DENV-2: number analyzed (Participants) | 1023 | 2049
  Year 3: DENV-2 | 73.5 | 99.9
  Year 3: DENV-3: number analyzed (Participants) | 1023 | 2049
  Year 3: DENV-3 | 70.2 | 95.7
  Year 3: DENV-4: number analyzed (Participants) | 1023 | 2049
  Year 3: DENV-4 | 71.1 | 96.0

13. Secondary Outcome: Seropositivity Rate for Multiple Dengue Serotypes in the Immunogenicity Subset
Description: Seropositivity rate for multiple Dengue serotypes, defined as the percentage of participants seropositive for any one (monovalent), two (bivalent), three (trivalent), and four (tetravalent) dengue serotypes, as well as at least bivalent (seropositive for ≥2 dengue serotypes) and at least trivalent (seropositive for ≥3 dengue serotypes), is derived from the titers of dengue-neutralizing antibodies. Seropositive response is defined as a reciprocal neutralizing titer ≥ 10. The four DENV serotypes are DENV-1, DENV-2, DENV-3 and DENV-4. Percentages were rounded off to the nearest single decimal place except the data points where rounding-up may lead to data misinterpretation.
Time Frame: as for outcome 12
Population: PPSI: all participants in FASI who had no major protocol violations. The FASI were based on FAS & included all randomized participants in subset for whom a valid pre-dosing and at least one valid post-dosing blood sample have been received for immunogenicity. Number analyzed is the number of participants with data available for analysis at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TDV 0.5 mL
Number analyzed (Participants) | 1247 | 2518
percentage of participants
  Baseline: Monovalent | 5.5 | 6.6
  Baseline: Bivalent | 3.8 | 2.4
  Baseline: Trivalent: number analyzed (Participants) | 1247 | 2517
  Baseline: Trivalent | 2.7 | 2.9
  Baseline: Tetravalent: number analyzed (Participants) | 1247 | 2517
  Baseline: Tetravalent | 60.4 | 60.2
  Baseline: At Least Bivalent | 66.9 | 65.5
  Baseline: At Least Trivalent: number analyzed (Participants) | 1247 | 2517
  Baseline: At Least Trivalent | 63.1 | 63.1
  Month 1: Monovalent: number analyzed (Participants) | 1165 | 2353
  Month 1: Monovalent | 7.4 | 0.3
  Month 1: Bivalent: number analyzed (Participants) | 1165 | 2353
  Month 1: Bivalent | 2.8 | 0.6
  Month 1: Trivalent: number analyzed (Participants) | 1164 | 2353
  Month 1: Trivalent | 3.2 | 3.7
  Month 1: Tetravalent: number analyzed (Participants) | 1164 | 2353
  Month 1: Tetravalent | 59.8 | 95.2
  Month 1: At Least Bivalent: number analyzed (Participants) | 1165 | 2353
  Month 1: At Least Bivalent | 65.8 | 99.4
  Month 1: At Least Trivalent: number analyzed (Participants) | 1164 | 2353
  Month 1: At Least Trivalent | 63.0 | 98.9
  Month 3: Monovalent: number analyzed (Participants) | 1244 | 2515
  Month 3: Monovalent | 6.8 | 0.4
  Month 3: Bivalent: number analyzed (Participants) | 1244 | 2515
  Month 3: Bivalent | 3.1 | 1.1
  Month 3: Trivalent: number analyzed (Participants) | 1244 | 2515
  Month 3: Trivalent | 3.1 | 3.7
  Month 3: Tetravalent: number analyzed (Participants) | 1243 | 2515
  Month 3: Tetravalent | 60.8 | 94.6
  Month 3: At Least Bivalent: number analyzed (Participants) | 1244 | 2515
  Month 3: At Least Bivalent | 67.0 | 99.4
  Month 3: At Least Trivalent: number analyzed (Participants) | 1244 | 2515
  Month 3: At Least Trivalent | 63.8 | 98.3
  Month 4: Monovalent: number analyzed (Participants) | 1131 | 2262
  Month 4: Monovalent | 6.6 | 0
  Month 4: Bivalent: number analyzed (Participants) | 1131 | 2262
  Month 4: Bivalent | 2.6 | 0.088
  Month 4: Trivalent: number analyzed (Participants) | 1131 | 2262
  Month 4: Trivalent | 2.5 | 0.1
  Month 4: Tetravalent: number analyzed (Participants) | 1131 | 2262
  Month 4: Tetravalent | 62.6 | 99.7
  Month 4: At Least Bivalent: number analyzed (Participants) | 1131 | 2262
  Month 4: At Least Bivalent | 67.6 | 99.956
  Month 4: At Least Trivalent: number analyzed (Participants) | 1131 | 2262
  Month 4: At Least Trivalent | 65.1 | 99.9
  Month 9: Monovalent: number analyzed (Participants) | 1085 | 2196
  Month 9: Monovalent | 7.7 | 0.091
  Month 9: Bivalent: number analyzed (Participants) | 1085 | 2196
  Month 9: Bivalent | 3.4 | 0.8
  Month 9: Trivalent: number analyzed (Participants) | 1085 | 2196
  Month 9: Trivalent | 2.0 | 2.1
  Month 9: Tetravalent: number analyzed (Participants) | 1085 | 2196
  Month 9: Tetravalent | 62.7 | 97.0
  Month 9: At Least Bivalent: number analyzed (Participants) | 1085 | 2196
  Month 9: At Least Bivalent | 68.1 | 99.909
  Month 9: At Least Trivalent: number analyzed (Participants) | 1085 | 2196
  Month 9: At Least Trivalent | 64.7 | 99.1
  Month 15: Monovalent: number analyzed (Participants) | 1115 | 2215
  Month 15: Monovalent | 3.9 | 0.5
  Month 15: Bivalent: number analyzed (Participants) | 1115 | 2215
  Month 15: Bivalent | 3.6 | 1.4
  Month 15: Trivalent: number analyzed (Participants) | 1115 | 2214
  Month 15: Trivalent | 2.1 | 2.2
  Month 15: Tetravalent: number analyzed (Participants) | 1115 | 2213
  Month 15: Tetravalent | 62.8 | 96.0
  Month 15: At Least Bivalent: number analyzed (Participants) | 1115 | 2215
  Month 15: At Least Bivalent | 68.4 | 99.5
  Month 15: At Least Trivalent: number analyzed (Participants) | 1115 | 2214
  Month 15: At Least Trivalent | 64.8 | 98.1
  Year 1: Monovalent: number analyzed (Participants) | 942 | 1904
  Year 1: Monovalent | 3.5 | 0.7
  Year 1: Bivalent: number analyzed (Participants) | 942 | 1904
  Year 1: Bivalent | 1.9 | 1.5
  Year 1: Trivalent: number analyzed (Participants) | 942 | 1904
  Year 1: Trivalent | 2.2 | 2.2
  Year 1: Tetravalent: number analyzed (Participants) | 942 | 1904
  Year 1: Tetravalent | 65.9 | 95.5
  Year 1: At Least Bivalent: number analyzed (Participants) | 942 | 1904
  Year 1: At Least Bivalent | 70.1 | 99.3
  Year 1: At Least Trivalent: number analyzed (Participants) | 942 | 1904
  Year 1: At Least Trivalent | 68.2 | 97.7
  Year 2: Monovalent: number analyzed (Participants) | 955 | 1921
  Year 2: Monovalent | 2.9 | 1.1
  Year 2: Bivalent: number analyzed (Participants) | 955 | 1921
  Year 2: Bivalent | 2.5 | 1.9
  Year 2: Trivalent: number analyzed (Participants) | 955 | 1921
  Year 2: Trivalent | 1.8 | 3.7
  Year 2: Tetravalent: number analyzed (Participants) | 955 | 1921
  Year 2: Tetravalent | 67.9 | 93.3
  Year 2: At Least Bivalent: number analyzed (Participants) | 955 | 1921
  Year 2: At Least Bivalent | 72.1 | 98.9
  Year 2: At Least Trivalent: number analyzed (Participants) | 955 | 1921
  Year 2: At Least Trivalent | 69.6 | 97.0
  Year 3:Monovalent: number analyzed (Participants) | 1023 | 2049
  Year 3:Monovalent | 2.6 | 1.6
  Year 3: Bivalent: number analyzed (Participants) | 1023 | 2049
  Year 3: Bivalent | 1.9 | 2.4
  Year 3:Trivalent: number analyzed (Participants) | 1023 | 2049
  Year 3:Trivalent | 2.5 | 3.7
  Year 3:Tetravalent: number analyzed (Participants) | 1023 | 2049
  Year 3:Tetravalent | 68.3 | 92.3
  Year 3:At Least Bivalent: number analyzed (Participants) | 1023 | 2049
  Year 3:At Least Bivalent | 72.7 | 98.3
  Year 3:At Least Trivalent: number analyzed (Participants) | 1023 | 2049
  Year 3:At Least Trivalent | 70.9 | 95.9

14. Secondary Outcome: Geometric Mean Titers (GMTs) of Neutralizing Antibodies for Each of the Four Dengue Serotypes in the Immunogenicity Subset
Description: GMTs of neutralizing antibodies were measured via microneutralization test 50% (MNT50). The four DENV serotypes are DENV-1, DENV-2, DENV-3 and DENV-4.
Time Frame: as for outcome 12
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: titres
Arm/Group | Placebo | TDV 0.5 mL
Number analyzed (Participants) | 1247 | 2518
titres
  Baseline: DENV-1 | 128.6 [109.3 to 151.4] | 120.3 [107.3 to 134.8]
  Baseline: DENV-2: number analyzed (Participants) | 1247 | 2517
  Baseline: DENV-2 | 197.4 [167.8 to 232.2] | 186.0 [165.9 to 208.4]
  Baseline: DENV-3: number analyzed (Participants) | 1247 | 2517
  Baseline: DENV-3 | 109.4 [93.8 to 127.6] | 108.7 [97.6 to 121.1]
  Baseline: DENV-4 | 80.8 [70.2 to 93.1] | 76.2 [69.2 to 83.9]
  Month 1: DENV-1: number analyzed (Participants) | 1165 | 2353
  Month 1: DENV-1 | 127.5 [107.7 to 150.9] | 1031.5 [944.4 to 1126.6]
  Month 1: DENV-2: number analyzed (Participants) | 1164 | 2353
  Month 1: DENV-2 | 197.2 [166.7 to 233.4] | 6575.7 [6237.2 to 6932.5]
  Month 1: DENV-3: number analyzed (Participants) | 1164 | 2353
  Month 1: DENV-3 | 108.6 [92.8 to 127.1] | 1133.8 [1050.4 to 1223.8]
  Month 1: DENV-4: number analyzed (Participants) | 1165 | 2353
  Month 1: DENV-4 | 77.6 [67.2 to 89.7] | 653.4 [607.0 to 703.4]
  Month 3: DENV-1: number analyzed (Participants) | 1244 | 2515
  Month 3: DENV-1 | 126.3 [107.9 to 148.0] | 828.7 [760.6 to 902.8]
  Month 3: DENV-2: number analyzed (Participants) | 1244 | 2515
  Month 3: DENV-2 | 201.0 [171.3 to 236.0] | 3598.5 [3425.0 to 3780.8]
  Month 3: DENV-3: number analyzed (Participants) | 1243 | 2515
  Month 3: DENV-3 | 103.9 [89.5 to 120.7] | 714.2 [661.1 to 771.6]
  Month 3: DENV-4: number analyzed (Participants) | 1244 | 2515
  Month 3: DENV-4 | 77.8 [67.8 to 89.3] | 463.9 [431.3 to 498.9]
  Month 4: DENV-1: number analyzed (Participants) | 1131 | 2262
  Month 4: DENV-1 | 139.0 [117.6 to 164.3] | 1059.2 [981.6 to 1143.0]
  Month 4: DENV-2: number analyzed (Participants) | 1131 | 2262
  Month 4: DENV-2 | 215.3 [181.7 to 255.0] | 3646.7 [3480.0 to 3821.3]
  Month 4: DENV-3: number analyzed (Participants) | 1131 | 2262
  Month 4: DENV-3 | 114.5 [97.7 to 134.3] | 986.7 [924.5 to 1053.0]
  Month 4: DENV-4: number analyzed (Participants) | 1131 | 2262
  Month 4: DENV-4 | 86.2 [74.5 to 99.8] | 630.0 [593.2 to 668.9]
  Month 9: DENV-1: number analyzed (Participants) | 1085 | 2196
  Month 9: DENV-1 | 130.5 [110.3 to 154.4] | 666.6 [611.8 to 726.2]
  Month 9: DENV-2: number analyzed (Participants) | 1085 | 2196
  Month 9: DENV-2 | 225.7 [190.5 to 267.3] | 2521.0 [2392.4 to 2656.5]
  Month 9: DENV-3: number analyzed (Participants) | 1085 | 2196
  Month 9: DENV-3 | 105.3 [89.9 to 123.3] | 513.0 [474.2 to 555.1]
  Month 9: DENV-4: number analyzed (Participants) | 1085 | 2196
  Month 9: DENV-4 | 84.4 [72.9 to 97.8] | 390.0 [363.6 to 418.4]
  Month 15: DENV-1: number analyzed (Participants) | 1115 | 2213
  Month 15: DENV-1 | 139.2 [117.6 to 164.7] | 584.1 [534.9 to 637.8]
  Month 15: DENV-2: number analyzed (Participants) | 1115 | 2214
  Month 15: DENV-2 | 211.8 [178.5 to 251.3] | 1977.3 [1871.7 to 2088.8]
  Month 15: DENV-3: number analyzed (Participants) | 1115 | 2215
  Month 15: DENV-3 | 97.3 [83.3 to 113.5] | 383.9 [354.0 to 416.3]
  Month 15: DENV-4: number analyzed (Participants) | 1115 | 2215
  Month 15: DENV-4 | 99.9 [86.0 to 116.0] | 408.0 [379.6 to 438.6]
  Year 1: DENV-1: number analyzed (Participants) | 942 | 1904
  Year 1: DENV-1 | 161.3 [134.6 to 193.3] | 567.8 [516.0 to 624.7]
  Year 1: DENV-2: number analyzed (Participants) | 942 | 1904
  Year 1: DENV-2 | 183.1 [154.0 to 217.7] | 1123.9 [1054.1 to 1198.3]
  Year 1: DENV-3: number analyzed (Participants) | 942 | 1904
  Year 1: DENV-3 | 111.0 [94.1 to 130.9] | 377.7 [346.2 to 412.2]
  Year 1: DENV-4: number analyzed (Participants) | 942 | 1904
  Year 1: DENV-4 | 98.6 [84.6 to 115.0] | 345.0 [319.6 to 372.5]
  Year 2: DENV-1: number analyzed (Participants) | 955 | 1921
  Year 2: DENV-1 | 205.1 [170.9 to 246.1] | 513.2 [465.9 to 565.3]
  Year 2: DENV-2: number analyzed (Participants) | 955 | 1921
  Year 2: DENV-2 | 208.1 [175.3 to 246.9] | 896.4 [839.2 to 957.5]
  Year 2: DENV-3: number analyzed (Participants) | 955 | 1921
  Year 2: DENV-3 | 127.5 [108.2 to 150.2] | 323.2 [295.7 to 353.2]
  Year 2: DENV-4: number analyzed (Participants) | 955 | 1921
  Year 2: DENV-4 | 110.4 [94.8 to 128.4] | 283.8 [262.9 to 306.4]
  Year 3: DENV-1: number analyzed (Participants) | 1023 | 2049
  Year 3: DENV-1 | 213.3 [179.4 to 253.6] | 483.1 [440.7 to 529.7]
  Year 3: DENV-2: number analyzed (Participants) | 1023 | 2049
  Year 3: DENV-2 | 193.6 [164.6 to 227.6] | 727.5 [682.4 to 775.5]
  Year 3: DENV-3: number analyzed (Participants) | 1023 | 2049
  Year 3: DENV-3 | 139.8 [119.3 to 163.7] | 327.9 [301.4 to 356.8]
  Year 3: DENV-4: number analyzed (Participants) | 1023 | 2049
  Year 3: DENV-4 | 107.6 [93.1 to 124.4] | 244.4 [226.7 to 263.6]

15. Other Pre Specified Outcome: VE of Two Doses of TDV in Preventing Virologically-Confirmed Dengue Fever Induced by Any Dengue Serotype
Description: VE is defined as 1 - (λv/λc), where λv and λc denote the hazard rates for the TDV and placebo arms, respectively. A virologically-confirmed dengue case is defined as febrile illness (defined as temperature ≥38°C on any 2 of 3 consecutive days) or illness clinically suspected to be dengue by the Investigator with a positive serotype-specific RT-PCR. VE was assessed using the number of cases due to virologically-confirmed dengue fever that occurred during the first half of Part 3.
Time Frame: First half of Part 3 (18 months beginning at Month 22)
Population: as for outcome 1
Measure: Number; unit: number of cases
Arm/Group | Placebo | TDV 0.5 mL
Number analyzed (Participants) | 6236 | 12510
number of cases | 228 | 252
Statistical Analysis 1: Comparison: Placebo vs TDV 0.5 mL; Test type: Other; Cox Proportional Hazard Model; VE = 47.4, 95% CI 2-sided [37.1 to 56.0] — [estimate comment as in outcome 3, analysis 1]

16. Other Pre Specified Outcome: VE of Two Doses of TDV in Preventing Virologically-Confirmed Dengue Fever Induced by Any Dengue Serotype
Description: VE is defined as 1 - (λv/λc), where λv and λc denote the hazard rates for the TDV and placebo arms, respectively. A virologically-confirmed dengue case is defined as febrile illness (defined as temperature ≥38°C on any 2 of 3 consecutive days) or illness clinically suspected to be dengue by the Investigator with a positive serotype-specific RT-PCR. VE was assessed using the number of cases due to virologically-confirmed dengue fever that occurred during the second half of Part 3.
Time Frame: Second half of Part 3 (18 months beginning at Month 40)
Population: as for outcome 1
Measure: Number; unit: number of cases
Arm/Group | Placebo | TDV 0.5 mL
Number analyzed (Participants) | 6102 | 12224
number of cases | 52 | 49
Statistical Analysis 1: Comparison: Placebo vs TDV 0.5 mL; Test type: Other; Cox Proportional Hazard Model; VE = 55.7, 95% CI 2-sided [34.5 to 70.0] — [estimate comment as in outcome 3, analysis 1]

17. Other Pre Specified Outcome: VE of Two Doses of TDV in Preventing Hospitalization Due to Virologically-Confirmed Dengue Fever Induced by Any Dengue Serotype
Description: VE is defined as 1 - (λv/λc), where λv and λc denote the hazard rates for the TDV and placebo arms, respectively. A virologically-confirmed dengue case is defined as febrile illness (defined as temperature ≥38°C on any 2 of 3 consecutive days) or illness clinically suspected to be dengue by the Investigator with a positive serotype-specific RT-PCR. VE was assessed using the number of cases requiring hospitalization due to virologically-confirmed dengue fever that occurred during the first half of Part 3.
Time Frame: First half of Part 3 (18 months beginning at Month 22)
Population: as for outcome 1
Measure: Number; unit: number of cases
Arm/Group | Placebo | TDV 0.5 mL
Number analyzed (Participants) | 6236 | 12510
number of cases | 43 | 24
Statistical Analysis 1: Comparison: Placebo vs TDV 0.5 mL; Test type: Other; Cox Proportional Hazard Model; VE = 73.5, 95% CI 2-sided [56.3 to 83.9] — [estimate comment as in outcome 3, analysis 1]

18. Other Pre Specified Outcome: VE of Two Doses of TDV in Preventing Hospitalization Due to Virologically-Confirmed Dengue Fever Induced by Any Dengue Serotype
Description: VE is defined as 1 - (λv/λc), where λv and λc denote the hazard rates for the TDV and placebo arms, respectively. A virologically-confirmed dengue case is defined as febrile illness (defined as temperature ≥38°C on any 2 of 3 consecutive days) or illness clinically suspected to be dengue by the Investigator with a positive serotype-specific RT-PCR. VE was assessed using the number of cases requiring hospitalization due to virologically-confirmed dengue fever that occurred during the second half of Part 3.
Time Frame: Second half of Part 3 (18 months beginning at Month 40)
Population: as for outcome 1
Measure: Number; unit: number of cases
Arm/Group | Placebo | TDV 0.5 mL
Number analyzed (Participants) | 6102 | 12224
number of cases | 15 | 2
Statistical Analysis 1: Comparison: Placebo vs TDV 0.5 mL; Test type: Other; Cox Proportional Hazard Model; VE = 93.7, 95% CI 2-sided [72.4 to 98.6] — [estimate comment as in outcome 3, analysis 1]

19. Other Pre Specified Outcome: VE of a TDV Booster Dose in Preventing Virologically-Confirmed Dengue Fever Induced by Any Dengue Serotype From 30 Days Post-Booster Vaccination (Day 30 Booster [b] (Month 1b)) Until the End of Part 4
Description: The VE is defined as 1 - (λv/λc), where λv and λc denote the hazard rates for the TDV and placebo arms, respectively. A virologically-confirmed dengue case is defined as febrile illness (defined as temperature ≥38°C on any 2 of 3 consecutive days) or illness clinically suspected to be dengue by the Investigator with a positive serotype-specific RT-PCR. VE was assessed using the number of virologically-confirmed dengue fever cases.
Time Frame: From 30 days post-booster vaccination (Day 30 booster [b] (Month 1b)) until the end of Part 4 (Month 13b)
Population: The Per-Protocol Set-Booster (PPS-B) included all participants in the FAS-B who had no major protocol violations. The Full Analysis Set-Booster (FAS-B) included all participants 4 to 11 years of age at the time of randomization in the trial (Day 1 [Month 0]) who were included in the PPS and who received the booster dose of trial vaccine (TDV or placebo).
Measure: Number; unit: number of cases
Arm/Group | Placebo | TDV 0.5 mL
Number analyzed (Participants) | 2981 | 5966
number of cases | 93 | 39
Statistical Analysis 1: Comparison: Placebo vs TDV 0.5 mL; Test type: Other; Cox Proportional Hazard Model; VE = 79.4, 95% CI 2-sided [70.1 to 85.9] — [estimate comment as in outcome 1, analysis 1]

20. Other Pre Specified Outcome: VE of a TDV Booster Dose in Preventing Virologically Confirmed Dengue Fever Induced by Each Dengue Serotype From 30 Days Post-Booster Vaccination (Day 30b [Month 1b]) Until the End of Part 4
Description: VE is defined as 1 - (λv/λc), where λv and λc denote the hazard rates for the TDV and placebo arms, respectively. A virologically-confirmed dengue case is defined as febrile illness (defined as temperature ≥38°C on any 2 of 3 consecutive days) or illness clinically suspected to be dengue by the Investigator with a positive serotype-specific RT-PCR. VE was assessed using the number of virologically-confirmed dengue fever cases.
Time Frame: From 30 days post-booster vaccination (Day 30b [Month 1b]) until the end of Part 4 (Month 13b)
Population: The PPS-B included all participants in the FAS-B who had no major protocol violations. The FAS-B included all participants 4 to 11 years of age at the time of randomization in the trial (Day 1 [Month 0]) who were included in the PPS and who received the booster dose of trial vaccine (TDV or placebo).
Measure: Number; unit: number of cases
Arm/Group | Placebo | TDV 0.5 mL
Number analyzed (Participants) | 2981 | 5966
number of cases
  DENV-1 | 32 | 15
  DENV-2 | 31 | 9
  DENV-3 | 4 | 3
  DENV-4 | 26 | 12
Statistical Analysis 1: Comparison: Placebo vs TDV 0.5 mL; DENV-1; Test type: Other; Cox Proportional Hazard Model; VE = 76.8, 95% CI 2-sided [57.1 to 87.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs TDV 0.5 mL; DENV-2; Test type: Other; Cox Proportional Hazard Model; VE = 85.7, 95% CI 2-sided [69.9 to 93.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs TDV 0.5 mL; DENV-3; Test type: Other; Cox Proportional Hazard Model; VE = 62, 95% CI 2-sided [-69.7 to 91.5] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs TDV 0.5 mL; DENV-4; Test type: Other; Cox Proportional Hazard Model; VE = 77.2, 95% CI 2-sided [54.8 to 88.5] — [estimate comment as in outcome 1, analysis 1]

21. Other Pre Specified Outcome: VE of a TDV Booster Dose in Preventing Virologically Confirmed Dengue Fever Induced by Any And Each Dengue Serotype in Dengue Seronegative Participants at Baseline From 30 Days Post-Booster Vaccination (Day 30b [Month 1b]) Until the End of Part 4
Description: VE is defined as 1 - (λv/λc), where λv and λc denote the hazard rates for the TDV and placebo arms, respectively. A virologically-confirmed dengue case is defined as febrile illness (defined as temperature ≥38°C on any 2 of 3 consecutive days) or illness clinically suspected to be dengue by the Investigator with a positive serotype-specific RT-PCR. VE was assessed using the number of virologically-confirmed dengue fever cases. Participants are counted only once for the "Any Dengue Serotype" category but counted separately for each dengue serotype they belong to.
Time Frame: From 30 days post-booster vaccination (Day 30b [Month 1b]) until the end of Part 4 (Month 13b)
Population: The PPS-B included all participants in the FAS-B who had no major protocol violations. The FAS-B included all participants 4 to 11 years of age at the time of randomization in the trial (Day 1 [Month 0]) who were included in the PPS and who received the booster dose of trial vaccine (TDV or placebo). Overall number of participants analyzed is the number of participants with seronegative baseline status and with data available for analyses.
Measure: Number; unit: number of cases
Arm/Group | Placebo | TDV 0.5 mL
Number analyzed (Participants) | 986 | 1928
number of cases
  Any Dengue Serotype | 26 | 11
  DENV-1 | 14 | 4
  DENV-2 | 5 | 1
  DENV-3 | 2 | 2
  DENV-4 | 5 | 4
Statistical Analysis 1: Comparison: Placebo vs TDV 0.5 mL; Any Dengue Serotype; Test type: Other; Cox Proportional Hazard Model; VE = 79.2, 95% CI 2-sided [57.8 to 89.7] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs TDV 0.5 mL; DENV-1; Test type: Other; Cox Proportional Hazard Model; VE = 86, 95% CI 2-sided [57.6 to 95.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs TDV 0.5 mL; DENV-2; Test type: Other; Cox Proportional Hazard Model; VE = 89.9, 95% CI 2-sided [13.5 to 98.8] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs TDV 0.5 mL; DENV-3; Test type: Other; Cox Proportional Hazard Model; VE = 42.7, 95% CI 2-sided [-307.5 to 92.0] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs TDV 0.5 mL; DENV-4; Test type: Other; Cox Proportional Hazard Model; VE = 61, 95% CI 2-sided [-45.1 to 89.5] — [estimate comment as in outcome 1, analysis 1]

22. Other Pre Specified Outcome: VE of a TDV Booster Dose in Preventing Virologically Confirmed Dengue Fever Induced by Any and Each Dengue Serotype in Dengue Seropositive Participants at Baseline From 30 Days Post-Booster Vaccination (Day 30b [Month 1b]) Until the End of Part 4
Description: as for outcome 21
Time Frame: From 30 days post-booster vaccination (Day 30b [Month 1b]) until the end of Part 4 (Month 13b)
Population: The PPS-B included all participants in the FAS-B who had no major protocol violations. The FAS-B included all participants 4 to 11 years of age at the time of randomization in the trial (Day 1 [Month 0]) who were included in the PPS and who received the booster dose of trial vaccine (TDV or placebo). Overall number of participants analyzed is the number of participants with seropositive baseline status and with data available for analyses.
Measure: Number; unit: number of cases
Arm/Group | Placebo | TDV 0.5 mL
Number analyzed (Participants) | 1995 | 4036
number of cases
  Any Dengue Serotype | 67 | 28
  DENV-1 | 18 | 11
  DENV-2 | 26 | 8
  DENV-3 | 2 | 1
  DENV-4 | 21 | 8
Statistical Analysis 1: Comparison: Placebo vs TDV 0.5 mL; Any Dengue Serotype; Test type: Other; Cox Proportional Hazard Model; VE = 79.6, 95% CI 2-sided [68.3 to 86.9] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs TDV 0.5 mL; DENV-1; Test type: Other; Cox Proportional Hazard Model; VE = 69.9, 95% CI 2-sided [36.4 to 85.8] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs TDV 0.5 mL; DENV-2; Test type: Other; Cox Proportional Hazard Model; VE = 84.9, 95% CI 2-sided [66.6 to 93.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs TDV 0.5 mL; DENV-3; Test type: Other; Cox Proportional Hazard Model; VE = 75.6, 95% CI 2-sided [-168.8 to 97.8] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs TDV 0.5 mL; Test type: Other; Cox Proportional Hazard Model; VE = 81, 95% CI 2-sided [57.2 to 91.6] — [estimate comment as in outcome 1, analysis 1]

23. Other Pre Specified Outcome: VE of a TDV Booster Dose in Preventing Hospitalization Due to Virologically Confirmed Dengue Fever Induced by Any Dengue Serotype From 30 Days Post-Booster Vaccination (Day 30b [Month 1b]) Until the End of Part 4
Description: VE is defined as 1 - (λv/λc), where λv and λc denote the hazard rates for the TDV and placebo arms, respectively. A virologically-confirmed dengue case is defined as febrile illness (defined as temperature ≥38°C on any 2 of 3 consecutive days) or illness clinically suspected to be dengue by the Investigator with a positive serotype-specific RT-PCR. VE was assessed using the number of cases requiring hospitalization due to virologically-confirmed dengue fever.
Time Frame: From 30 days post-booster vaccination (Day 30b [Month 1b]) until the end of Part 4 (Month 13b)
Population: as for outcome 20
Measure: Number; unit: number of cases
Arm/Group | Placebo | TDV 0.5 mL
Number analyzed (Participants) | 2981 | 5966
number of cases | 24 | 3
Statistical Analysis 1: Comparison: Placebo vs TDV 0.5 mL; Test type: Other; Cox Proportional Hazard Model; VE = 93.8, 95% CI 2-sided [79.3 to 98.1] — [estimate comment as in outcome 3, analysis 1]

24. Other Pre Specified Outcome: VE of a TDV Booster Dose in Preventing Virologically Confirmed Severe Dengue Fever Induced by Any Dengue Serotype From 30 Days Post-Booster Vaccination (Day 30b [Month 1b]) Until the End of Part 4
Description: VE is defined as 1 - (λv/λc), where λv and λc denote the hazard rates for the TDV and placebo arms, respectively. A virologically-confirmed dengue case is defined as febrile illness (defined as temperature ≥38°C on any 2 of 3 consecutive days) or illness clinically suspected to be dengue by the Investigator with a positive serotype-specific RT-PCR. Severe cases were determined by Adjudication Committee. VE was assessed using the number of severe cases due to virologically-confirmed dengue fever.
Time Frame: From 30 days post-booster vaccination (Day 30b [Month 1b]) until the end of Part 4 (Month 13b)
Population: as for outcome 20
Measure: Number; unit: number of cases
Arm/Group | Placebo | TDV 0.5 mL
Number analyzed (Participants) | 2981 | 5966
number of cases | 1 | 0
Statistical Analysis 1: Comparison: Placebo vs TDV 0.5 mL; Test type: Other; Cox Proportional Hazard Model; VE = 100, 95% CI 2-sided [-849.4 to 100.0] — [estimate comment as in outcome 1, analysis 1]

25. Other Pre Specified Outcome: VE of a TDV Booster Dose in Preventing Virologically-Confirmed Dengue Fever Induced by Any Dengue Serotype During Part 5
Description: The VE is defined as 1 - (λv/λc), where λv and λc denote the hazard rates for the TDV and placebo arms, respectively. A virologically-confirmed dengue case is defined as febrile illness (defined as temperature ≥38°C on any 2 of 3 consecutive days) or illness clinically suspected to be dengue by the Investigator with a positive serotype-specific RT-PCR. VE was assessed using the number of virologically-confirmed dengue fever cases. Participants are counted only once for the any dengue serotype.
Time Frame: From Month 14b until the end of Part 5 (Month 25b)
Population: as for outcome 19
Measure: Number; unit: number of cases
Arm/Group | Placebo | TDV 0.5 mL
Number analyzed (Participants) | 2935 | 5865
number of cases | 66 | 45
Statistical Analysis 1: Comparison: Placebo vs TDV 0.5 mL; Test type: Other; Cox Proportional Hazard Model; VE = 67.2, 95% CI 2-sided [52.1 to 77.5] — [estimate comment as in outcome 1, analysis 1]

26. Other Pre Specified Outcome: VE of a TDV Booster Dose in Preventing Virologically Confirmed Dengue Fever Induced by Each Dengue Serotype During Part 5
Description: VE is defined as 1 - (λv/λc), where λv and λc denote the hazard rates for the TDV and placebo arms, respectively. A virologically-confirmed dengue case is defined as febrile illness (defined as temperature ≥38°C on any 2 of 3 consecutive days) or illness clinically suspected to be dengue by the Investigator with a positive serotype-specific RT-PCR. VE was assessed using the number of virologically-confirmed dengue fever cases. Participants are counted separately for each dengue serotype.
Time Frame: From Month 14b until the end of Part 5 (Month 25b)
Population: as for outcome 20
Measure: Number; unit: number of cases
Arm/Group | Placebo | TDV 0.5 mL
Number analyzed (Participants) | 2935 | 5865
number of cases
  DENV-1 | 19 | 17
  DENV-2 | 18 | 5
  DENV-3 | 20 | 20
  DENV-4 | 10 | 3
Statistical Analysis 1: Comparison: Placebo vs TDV 0.5 mL; DENV-1; Test type: Other; Cox Proportional Hazard Model; VE = 56.5, 95% CI 2-sided [16.2 to 77.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs TDV 0.5 mL; DENV-2; Test type: Other; Cox Proportional Hazard Model; VE = 86.6, 95% CI 2-sided [63.8 to 95.0] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs TDV 0.5 mL; DENV-3; Test type: Other; Cox Proportional Hazard Model; VE = 51.5, 95% CI 2-sided [9.9 to 73.9] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs TDV 0.5 mL; DENV-4; Test type: Other; Cox Proportional Hazard Model; VE = 85.5, 95% CI 2-sided [47.4 to 96.0] — [estimate comment as in outcome 1, analysis 1]

27. Other Pre Specified Outcome: VE of a TDV Booster Dose in Preventing Virologically Confirmed Dengue Fever Induced by Any And Each Dengue Serotype in Dengue Seronegative Participants at Baseline During Part 5
Description: as for outcome 21
Time Frame: From Month 14b until the end of Part 5 (Month 25b)
Population: as for outcome 21
Measure: Number; unit: number of cases
Arm/Group | Placebo | TDV 0.5 mL
Number analyzed (Participants) | 974 | 1908
number of cases
  Any Dengue Serotype | 20 | 12
  DENV-1 | 7 | 6
  DENV-2 | 5 | 1
  DENV-3 | 4 | 5
  DENV-4 | 4 | 0
Statistical Analysis 1: Comparison: Placebo vs TDV 0.5 mL; Any Dengue Serotype; Test type: Other; Cox Proportional Hazard Model; VE = 70.3, 95% CI 2-sided [39.1 to 85.5] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs TDV 0.5 mL; DENV-1; Test type: Other; Cox Proportional Hazard Model; VE = 57.3, 95% CI 2-sided [-27.2 to 85.7] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs TDV 0.5 mL; DENV-2; Test type: Other; Cox Proportional Hazard Model; VE = 90, 95% CI 2-sided [14.0 to 98.8] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs TDV 0.5 mL; DENV-3; Test type: Other; Cox Proportional Hazard Model; VE = 36.1, 95% CI 2-sided [-138.1 to 82.9] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs TDV 0.5 mL; DENV-4; Test type: Other; Cox Proportional Hazard Model; VE = 100, 95% CI 2-sided [43.1 to 100.0] — [estimate comment as in outcome 1, analysis 1]

28. Other Pre Specified Outcome: VE of a TDV Booster Dose in Preventing Virologically Confirmed Dengue Fever Induced by Any and Each Dengue Serotype in Dengue Seropositive Participants at Baseline During Part 5
Description: as for outcome 21
Time Frame: From Month 14b until the end of Part 5 (Month 25b)
Population: as for outcome 22
Measure: Number; unit: number of cases
Arm/Group | Placebo | TDV 0.5 mL
Number analyzed (Participants) | 1961 | 3955
number of cases
  Any Dengue Serotype | 46 | 33
  DENV-1 | 12 | 11
  DENV-2 | 13 | 4
  DENV-3 | 16 | 15
  DENV-4 | 6 | 3
Statistical Analysis 1: Comparison: Placebo vs TDV 0.5 mL; Any Dengue Serotype; Test type: Other; Cox Proportional Hazard Model; VE = 65.7, 95% CI 2-sided [46.4 to 78.1] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs TDV 0.5 mL; DENV-1; Test type: Other; Cox Proportional Hazard Model; VE = 56.2, 95% CI 2-sided [0.8 to 80.7] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs TDV 0.5 mL; DENV-2; Test type: Other; Cox Proportional Hazard Model; VE = 85.1, 95% CI 2-sided [54.4 to 95.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs TDV 0.5 mL; DENV-3; Test type: Other; Cox Proportional Hazard Model; VE = 54.7, 95% CI 2-sided [8.3 to 77.6] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs TDV 0.5 mL; Test type: Other; Cox Proportional Hazard Model; VE = 75.5, 95% CI 2-sided [2.2 to 93.9] — [estimate comment as in outcome 1, analysis 1]

29. Other Pre Specified Outcome: VE of a TDV Booster Dose in Preventing Hospitalization Due to Virologically Confirmed Dengue Fever Induced by Any Dengue Serotype During Part 5
Description: as for outcome 23
Time Frame: From Month 14b until the end of Part 5 (Month 25b)
Population: as for outcome 20
Measure: Number; unit: number of cases
Arm/Group | Placebo | TDV 0.5 mL
Number analyzed (Participants) | 2935 | 5865
number of cases | 13 | 4
Statistical Analysis 1: Comparison: Placebo vs TDV 0.5 mL; Test type: Other; Cox Proportional Hazard Model; VE = 84.9, 95% CI 2-sided [53.7 to 95.1] — [estimate comment as in outcome 3, analysis 1]

30. Other Pre Specified Outcome: VE of a TDV Booster Dose in Preventing Virologically Confirmed Severe Dengue Fever Induced by Any Dengue Serotype During Part 5
Description: as for outcome 24
Time Frame: From Month 14b until the end of Part 5 (Month 25b)
Population: as for outcome 20
Measure: Number; unit: number of cases
Arm/Group | Placebo | TDV 0.5 mL
Number analyzed (Participants) | 2935 | 5865
number of cases | 0 | 0

31. Other Pre Specified Outcome: VE of a TDV Booster Dose in Preventing Virologically-Confirmed Dengue Fever Induced by Any Dengue Serotype for Parts 4 And 5 Combined
Description: as for outcome 19
Time Frame: From 30 days post-booster vaccination (Day 30b [Month 1b) until the end of Part 5 (Month 25b)
Population: as for outcome 20
Measure: Number; unit: number of cases
Arm/Group | Placebo | TDV 0.5 mL
Number analyzed (Participants) | 2981 | 5966
number of cases | 159 | 84
Statistical Analysis 1: Comparison: Placebo vs TDV 0.5 mL; Test type: Other; Cox Proportional Hazard Model; VE = 74.3, 95% CI 2-sided [66.6 to 80.3] — [estimate comment as in outcome 1, analysis 1]

32. Other Pre Specified Outcome: VE of a TDV Booster Dose in Preventing Virologically Confirmed Dengue Fever Induced by Each Dengue Serotype for Parts 4 And 5 Combined
Description: as for outcome 20
Time Frame: From 30 days post-booster vaccination (Day 30b [Month 1b]) until the end of Part 5 (Month 25b)
Population: as for outcome 20
Measure: Number; unit: number of cases
Arm/Group | Placebo | TDV 0.5 mL
Number analyzed (Participants) | 2981 | 5966
number of cases
  DENV-1 | 51 | 32
  DENV-2 | 49 | 14
  DENV-3 | 25 | 23
  DENV-4 | 36 | 15
Statistical Analysis 1: Comparison: Placebo vs TDV 0.5 mL; DENV-1; Test type: Other; Cox Proportional Hazard Model; VE = 69, 95% CI 2-sided [51.7 to 80.0] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs TDV 0.5 mL; DENV-2; Test type: Other; Cox Proportional Hazard Model; VE = 85.9, 95% CI 2-sided [74.5 to 92.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs TDV 0.5 mL; DENV-3; Test type: Other; Cox Proportional Hazard Model; VE = 54.1, 95% CI 2-sided [19.1 to 73.9] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs TDV 0.5 mL; DENV-4; Test type: Other; Cox Proportional Hazard Model; VE = 79.4, 95% CI 2-sided [62.4 to 88.7] — [estimate comment as in outcome 1, analysis 1]

33. Other Pre Specified Outcome: VE of a TDV Booster Dose in Preventing Virologically Confirmed Dengue Fever Induced by Any And Each Dengue Serotype in Dengue Seronegative Participants at Baseline for Parts 4 And 5 Combined
Description: as for outcome 21
Time Frame: From 30 days post-booster vaccination (Day 30b [Month 1b]) until the end of Part 5 (Month 25b)
Population: as for outcome 21
Measure: Number; unit: number of cases
Arm/Group | Placebo | TDV 0.5 mL
Number analyzed (Participants) | 986 | 1928
number of cases
  Any Dengue Serotype | 46 | 23
  DENV-1 | 21 | 10
  DENV-2 | 10 | 2
  DENV-3 | 6 | 7
  DENV-4 | 9 | 4
Statistical Analysis 1: Comparison: Placebo vs TDV 0.5 mL; Any Dengue Serotype; Test type: Other; Cox Proportional Hazard Model; VE = 75.3, 95% CI 2-sided [59.3 to 85.0] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs TDV 0.5 mL; DENV-1; Test type: Other; Cox Proportional Hazard Model; VE = 76.5, 95% CI 2-sided [50.0 to 88.9] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs TDV 0.5 mL; DENV-2; Test type: Other; Cox Proportional Hazard Model; VE = 89.9, 95% CI 2-sided [53.7 to 97.8] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs TDV 0.5 mL; DENV-3; Test type: Other; Cox Proportional Hazard Model; VE = 37.9, 95% CI 2-sided [-84.9 to 79.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs TDV 0.5 mL; DENV-4; Test type: Other; Cox Proportional Hazard Model; VE = 78.4, 95% CI 2-sided [29.7 to 93.3] — [estimate comment as in outcome 1, analysis 1]

34. Other Pre Specified Outcome: VE of a TDV Booster Dose in Preventing Virologically Confirmed Dengue Fever Induced by Any and Each Dengue Serotype in Dengue Seropositive Participants at Baseline for Parts 4 And 5 Combined
Description: as for outcome 21
Time Frame: From 30 days post-booster vaccination (Day 30b [Month 1b]) until the end of Part 5 (Month 25b)
Population: as for outcome 22
Measure: Number; unit: number of cases
Arm/Group | Placebo | TDV 0.5 mL
Number analyzed (Participants) | 1995 | 4036
number of cases
  Any Dengue Serotype | 113 | 61
  DENV-1 | 30 | 22
  DENV-2 | 39 | 12
  DENV-3 | 19 | 16
  DENV-4 | 27 | 11
Statistical Analysis 1: Comparison: Placebo vs TDV 0.5 mL; Any Dengue Serotype; Test type: Other; Cox Proportional Hazard Model; VE = 73.9, 95% CI 2-sided [64.4 to 80.9] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs TDV 0.5 mL; DENV-1; Test type: Other; Cox Proportional Hazard Model; VE = 64.1, 95% CI 2-sided [37.8 to 79.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs TDV 0.5 mL; DENV-2; Test type: Other; Cox Proportional Hazard Model; VE = 84.9, 95% CI 2-sided [71.1 to 92.1] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs TDV 0.5 mL; DENV-3; Test type: Other; Cox Proportional Hazard Model; VE = 58.1, 95% CI 2-sided [18.5 to 78.5] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs TDV 0.5 mL; Test type: Other; Cox Proportional Hazard Model; VE = 79.7, 95% CI 2-sided [59.1 to 89.9] — [estimate comment as in outcome 1, analysis 1]

35. Other Pre Specified Outcome: VE of a TDV Booster Dose in Preventing Hospitalization Due to Virologically Confirmed Dengue Fever Induced by Any Dengue Serotype for Parts 4 And 5 Combined
Description: as for outcome 23
Time Frame: From 30 days post-booster vaccination (Day 30b [Month 1b]) until the end of Part 5 (Month 25b)
Population: as for outcome 20
Measure: Number; unit: number of cases
Arm/Group | Placebo | TDV 0.5 mL
Number analyzed (Participants) | 2981 | 5966
number of cases | 37 | 7
Statistical Analysis 1: Comparison: Placebo vs TDV 0.5 mL; Test type: Other; Cox Proportional Hazard Model; VE = 90.6, 95% CI 2-sided [78.8 to 95.8] — [estimate comment as in outcome 3, analysis 1]

36. Other Pre Specified Outcome: VE of a TDV Booster Dose in Preventing Virologically Confirmed Severe Dengue Fever Induced by Any Dengue Serotype for Parts 4 And 5 Combined
Description: as for outcome 24
Time Frame: From 30 days post-booster vaccination (Day 30b [Month 1b]) until the end of Part 5 (Month 25b)
Population: as for outcome 20
Measure: Number; unit: number of cases
Arm/Group | Placebo | TDV 0.5 mL
Number analyzed (Participants) | 2981 | 5966
number of cases | 1 | 0
Statistical Analysis 1: Comparison: Placebo vs TDV 0.5 mL; Test type: Other; Cox Proportional Hazard Model; VE = 100, 95% CI 2-sided [-849.4 to 100.0] — [estimate comment as in outcome 3, analysis 1]

37. Other Pre Specified Outcome: Percentage of Participants With Solicited Local Injection Site Adverse Events (AEs) by Severity in the Safety Set-Booster-Immunogenicity Subset During Part 4
Description: Solicited local AEs at injection site are defined as pain, erythema and swelling that occurred within 7 days after each vaccination. The participant/legal guardian recorded the severity of each AE (except erythema and swelling) according to the diary card instruction as none, mild, moderate, or severe. Severity grades for erythema and swelling were derived from the recorded diameters. Percentages were rounded off to the nearest single decimal place.
Time Frame: Days 1b through 7b after booster vaccination in Part 4
Population: Safety Set-Booster-Immunogenicity Subset included all participants 4 to 11 years of age at the time of randomization in the trial (Day 1 [Month 0]) who were included in the PPS and who received the booster dose of trial vaccine (TDV or placebo) in the safety subset. Number analyzed is the number of participants with data available for analyses for the specified category.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TDV 0.5 mL
Number analyzed (Participants) | 600 | 1200
percentage of participants
  Pain: Mild: number analyzed (Participants) | 595 | 1182
  Pain: Mild | 12.1 | 20.1
  Pain: Moderate: number analyzed (Participants) | 595 | 1182
  Pain: Moderate | 3.9 | 4.6
  Pain: Severe: number analyzed (Participants) | 595 | 1182
  Pain: Severe | 0.7 | 1.2
  Erythema: Mild: number analyzed (Participants) | 592 | 1174
  Erythema: Mild | 0.2 | 1.6
  Erythema: Moderate: number analyzed (Participants) | 592 | 1174
  Erythema: Moderate | 0 | 0
  Erythema: Severe: number analyzed (Participants) | 592 | 1174
  Erythema: Severe | 0 | 0
  Swelling: Mild: number analyzed (Participants) | 590 | 1173
  Swelling: Mild | 0.5 | 1.0
  Swelling: Moderate: number analyzed (Participants) | 590 | 1173
  Swelling: Moderate | 0 | 0
  Swelling: Severe: number analyzed (Participants) | 590 | 1173
  Swelling: Severe | 0 | 0

38. Other Pre Specified Outcome: Percentage of Participants With Solicited Systemic Adverse Events (AEs) by Severity in the Safety Set-Booster-Immunogenicity Subset During Part 4
Description: Solicited systemic AEs are defined as fever, headache, asthenia, malaise and myalgia that occurred within 14 days after each vaccination. The participant/legal guardian recorded the severity of each AE (except fever) according to the diary card instruction as none, mild, moderate, or severe. Severity grades for fever were derived from the recorded body temperature measurements and presented using the proposed temperature increments published by the Brighton Collaboration. Percentages were rounded off to the nearest single decimal place except the data point where rounding-up may lead to data misinterpretation.
Time Frame: Days 1b through 14b after booster vaccination in Part 4
Population: as for outcome 37
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TDV 0.5 mL
Number analyzed (Participants) | 600 | 1200
percentage of participants
  Headache: Mild: number analyzed (Participants) | 594 | 1184
  Headache: Mild | 8.6 | 12.3
  Headache: Moderate: number analyzed (Participants) | 594 | 1184
  Headache: Moderate | 4.7 | 3.7
  Headache: Severe: number analyzed (Participants) | 594 | 1184
  Headache: Severe | 0.5 | 1.1
  Asthenia: Mild: number analyzed (Participants) | 594 | 1184
  Asthenia: Mild | 7.1 | 7.2
  Asthenia: Moderate: number analyzed (Participants) | 594 | 1184
  Asthenia: Moderate | 1.9 | 2.4
  Asthenia: Severe: number analyzed (Participants) | 594 | 1184
  Asthenia: Severe | 0.3 | 0.7
  Malaise: Mild: number analyzed (Participants) | 593 | 1184
  Malaise: Mild | 7.6 | 8.6
  Malaise: Moderate: number analyzed (Participants) | 593 | 1184
  Malaise: Moderate | 2.0 | 2.6
  Malaise: Severe: number analyzed (Participants) | 593 | 1184
  Malaise: Severe | 0.5 | 0.7
  Myalgia: Mild: number analyzed (Participants) | 593 | 1181
  Myalgia: Mild | 9.9 | 11.7
  Myalgia: Moderate: number analyzed (Participants) | 593 | 1181
  Myalgia: Moderate | 1.5 | 3.6
  Myalgia: Severe: number analyzed (Participants) | 593 | 1181
  Myalgia: Severe | 1.0 | 0.8
  Fever: 38.0-<38.5: number analyzed (Participants) | 584 | 1146
  Fever: 38.0-<38.5 | 1.0 | 1.8
  Fever: 38.5-<39.0: number analyzed (Participants) | 584 | 1146
  Fever: 38.5-<39.0 | 0.5 | 1.0
  Fever: 39.0-<39.5: number analyzed (Participants) | 584 | 1146
  Fever: 39.0-<39.5 | 0.2 | 0.2
  Fever: 39.5-<40.0: number analyzed (Participants) | 584 | 1146
  Fever: 39.5-<40.0 | 0 | 0.3
  Fever: 40.0-<40.5: number analyzed (Participants) | 584 | 1146
  Fever: 40.0-<40.5 | 0.2 | 0
  Fever: 40.5-<41.0: number analyzed (Participants) | 584 | 1146
  Fever: 40.5-<41.0 | 0 | 0.0873
  Fever: >=41.0: number analyzed (Participants) | 584 | 1146
  Fever: >=41.0 | 0 | 0

39. Other Pre Specified Outcome: Percentage of Participants With Any Unsolicited Adverse Events (AEs) in the Safety Set-Booster-Immunogenicity Subset During Part 4
Description: as for outcome 9
Time Frame: Days 1b through 28b after booster vaccination in Part 4
Population: Safety Set-Booster-Immunogenicity Subset included all participants 4 to 11 years of age at the time of randomization in the trial (Day 1 [Month 0]) who were included in the PPS and who received the booster dose of trial vaccine (TDV or placebo) in the safety subset.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TDV 0.5 mL
Number analyzed (Participants) | 600 | 1200
percentage of participants | 1.8 | 1.8

40. Other Pre Specified Outcome: Percentage of Participants With Serious Adverse Events (SAEs) During Parts 4 and 5
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a trial vaccine; it does not necessarily have to have a causal relationship with trial vaccine administration. A serious adverse event (SAE) is any untoward medical occurrence or effect that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability / incapacity, is a congenital anomaly / birth defect or is medically important due to other reasons than the above mentioned criteria. Percentages were rounded off to the nearest single decimal place. In the category 'Part 4 and 5 combined' participants are counted only once even if they experienced events in both Part 4 and Part 5 in order to yield total of unique participants who had SAEs.
Time Frame: From Day 1b until the end of Part 4 (Month 13b) and Part 5 (Month 25b)
Population: Safety Set-Booster (SS-B) included all participants 4 to 11 years of age at the time of randomization in the trial (Day 1 [Month 0]) who were included in the PPS and who received the booster dose of trial vaccine (TDV or placebo). Number analyzed is the number of participants at risk at the start of the specified analysis period.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TDV 0.5 mL
Number analyzed (Participants) | 2985 | 5990
percentage of participants
  Part 4 | 4.2 | 2.7
  Part 5: number analyzed (Participants) | 2939 | 5889
  Part 5 | 2.5 | 1.9
  Parts 4 and 5 Combined | 6.4 | 4.4

41. Other Pre Specified Outcome: Percentage of Participants With Fatal SAEs and SAEs Related to Study Drug During Parts 4 and 5
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a trial vaccine; it does not necessarily have to have a causal relationship with trial vaccine administration. A SAE is any untoward medical occurrence or effect that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability / incapacity, is a congenital anomaly / birth defect or is medically important due to other reasons than the above mentioned criteria. Percentages were rounded off to the nearest single decimal place except the data points where rounding-up may lead to data misinterpretation. In the category 'Part 4 and 5 combined' participants are counted only once even if they experienced events in both Part 4 and Part 5 in order to yield total of unique participants who had SAEs.
Time Frame: From Day 1b until the end of Part 4 (Month 13b) and Part 5 (Month 25b)
Population: SS-B included all participants 4 to 11 years of age at the time of randomization in the trial (Day 1 [Month 0]) who were included in the PPS and who received the booster dose of trial vaccine (TDV or placebo). Number analyzed is the number of participants at risk at the start of the specified analysis period.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TDV 0.5 mL
Number analyzed (Participants) | 2985 | 5990
percentage of participants
  Part 4: Fatal SAEs | 0.0335 | 0.0501
  Part 4: SAEs Related to Study Drug | 0 | 0
  Part 5: Fatal SAEs: number analyzed (Participants) | 2939 | 5889
  Part 5: Fatal SAEs | 0 | 0.0509
  Part 5: SAEs Related to Study Drug: number analyzed (Participants) | 2939 | 5889
  Part 5: SAEs Related to Study Drug | 0 | 0
  Parts 4&5 Combined: Fatal SAEs | 0.0335 | 0.1
  Parts 4&5 Combined: SAEs Related to Study Drug | 0 | 0

42. Other Pre Specified Outcome: Seropositivity Rate for Each of The 4 Dengue Serotypes During Parts 4 and 5
Description: as for outcome 12
Time Frame: Pre-booster Vaccination on Day 1b (Month 0b) and post-booster vaccination on Day 30b (Month 1b), Day 180b (Month 6b), Day 395b (Month 13b) and Day 760b (Month 25b) in Parts 4 and 5
Population: Per-Protocol Set for Immunogenicity-Booster (PPSI-B):all participants in Full Analysis Set for Immunogenicity-Booster (FASI-B) who had no major protocol violations. FASI-B: all participants from FAS-B who were included in booster immunogenicity subset & for whom there is valid pre-booster measurement & at least 1 valid post-booster measurement for immunogenicity assessments. Number analyzed: participants with data available for analyses for the specified category.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TDV 0.5 mL
Number analyzed (Participants) | 597 | 1186
percentage of participants
  Day 1b: DENV-1 | 70.2 | 94.4
  Day 1b: DENV-2 | 72.5 | 99.2
  Day 1b: DENV-3 | 69.0 | 97.0
  Day 1b: DENV-4 | 67.0 | 93.4
  Month 1b: DENV-1: number analyzed (Participants) | 542 | 1075
  Month 1b: DENV-1 | 71.6 | 99.907
  Month 1b: DENV-2: number analyzed (Participants) | 542 | 1075
  Month 1b: DENV-2 | 74.5 | 99.907
  Month 1b: DENV-3: number analyzed (Participants) | 542 | 1075
  Month 1b: DENV-3 | 72.9 | 100.0
  Month 1b: DENV-4: number analyzed (Participants) | 542 | 1075
  Month 1b: DENV-4 | 69.2 | 99.7
  Month 6b: DENV-1: number analyzed (Participants) | 562 | 1127
  Month 6b: DENV-1 | 72.8 | 99.7
  Month 6b: DENV-2: number analyzed (Participants) | 562 | 1126
  Month 6b: DENV-2 | 75.8 | 99.8
  Month 6b: DENV-3: number analyzed (Participants) | 562 | 1127
  Month 6b: DENV-3 | 73.0 | 99.6
  Month 6b: DENV-4: number analyzed (Participants) | 562 | 1127
  Month 6b: DENV-4 | 70.3 | 99.7
  Month 13b: DENV-1: number analyzed (Participants) | 561 | 1122
  Month 13b: DENV-1 | 74.5 | 99.911
  Month 13b: DENV-2: number analyzed (Participants) | 561 | 1122
  Month 13b: DENV-2 | 77.4 | 99.5
  Month 13b: DENV-3: number analyzed (Participants) | 561 | 1122
  Month 13b: DENV-3 | 74.9 | 100.0
  Month 13b: DENV-4: number analyzed (Participants) | 561 | 1122
  Month 13b: DENV-4 | 72.4 | 99.8
  Month 25b: DENV-1: number analyzed (Participants) | 556 | 1103
  Month 25b: DENV-1 | 77.2 | 99.6
  Month 25b: DENV-2: number analyzed (Participants) | 556 | 1103
  Month 25b: DENV-2 | 78.6 | 99.8
  Month 25b: DENV-3: number analyzed (Participants) | 556 | 1102
  Month 25b: DENV-3 | 77.7 | 99.909
  Month 25b: DENV-4: number analyzed (Participants) | 556 | 1103
  Month 25b: DENV-4 | 76.3 | 99.8

43. Other Pre Specified Outcome: Seropositivity Rate for Multiple Dengue Serotypes During Parts 4 and 5
Description: as for outcome 13
Time Frame: as for outcome 42
Population: PPSI-B: all participants in FASI-B who had no major protocol violations. FASI-B: all participants from FAS-B who were included in booster immunogenicity subset & for whom there is valid pre-booster measurement & at least 1 valid post-booster measurement for immunogenicity assessments. Number analyzed: number of participants with data available for analyses for specified category.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TDV 0.5 mL
Number analyzed (Participants) | 597 | 1186
percentage of participants
  Day 1b: Monovalent | 5.7 | 1.3
  Day 1b: Bivalent | 2.0 | 3.7
  Day 1b: Trivalent | 2.3 | 4.6
  Day 1b: Tetravalent | 65.5 | 90.4
  Day 1b: At Least Bivalent | 69.8 | 98.7
  Day 1b: At Least Trivalent | 67.8 | 95.0
  Month 1b: Monovalent: number analyzed (Participants) | 542 | 1075
  Month 1b: Monovalent | 6.6 | 0
  Month 1b: Bivalent: number analyzed (Participants) | 542 | 1075
  Month 1b: Bivalent | 2.0 | 0
  Month 1b: Trivalent: number analyzed (Participants) | 542 | 1075
  Month 1b: Trivalent | 3.7 | 0.5
  Month 1b: Tetravalent: number analyzed (Participants) | 542 | 1075
  Month 1b: Tetravalent | 66.6 | 99.5
  Month 1b:At Least Bivalent: number analyzed (Participants) | 542 | 1075
  Month 1b:At Least Bivalent | 72.3 | 100.0
  Month 1b:At Least Trivalent: number analyzed (Participants) | 542 | 1075
  Month 1b:At Least Trivalent | 70.3 | 100.0
  Month 6b:Monovalent: number analyzed (Participants) | 562 | 1127
  Month 6b:Monovalent | 6.8 | 0.0887
  Month 6b: Bivalent: number analyzed (Participants) | 562 | 1127
  Month 6b: Bivalent | 2.5 | 0.0887
  Month 6b: Trivalent: number analyzed (Participants) | 562 | 1127
  Month 6b: Trivalent | 3.2 | 0.6
  Month 6b: Tetravalent: number analyzed (Participants) | 562 | 1126
  Month 6b: Tetravalent | 67.6 | 99.2
  Month 6b:At Least Bivalent: number analyzed (Participants) | 562 | 1127
  Month 6b:At Least Bivalent | 73.3 | 99.911
  Month 6b:At Least Trivalent: number analyzed (Participants) | 562 | 1127
  Month 6b:At Least Trivalent | 70.8 | 99.8
  Month 13b: Monovalent: number analyzed (Participants) | 561 | 1122
  Month 13b: Monovalent | 6.6 | 0
  Month 13b: Bivalent: number analyzed (Participants) | 561 | 1122
  Month 13b: Bivalent | 2.1 | 0
  Month 13b: Trivalent: number analyzed (Participants) | 561 | 1122
  Month 13b: Trivalent | 2.7 | 0.8
  Month 13b: Tetravalent: number analyzed (Participants) | 561 | 1122
  Month 13b: Tetravalent | 70.1 | 99.2
  Month 13b: At Least Bivalent: number analyzed (Participants) | 561 | 1122
  Month 13b: At Least Bivalent | 74.9 | 100.0
  Month 13b: At Least Trivalent: number analyzed (Participants) | 561 | 1122
  Month 13b: At Least Trivalent | 72.7 | 100.0
  Month 25b: Monovalent: number analyzed (Participants) | 556 | 1103
  Month 25b: Monovalent | 3.4 | 0
  Month 25b: Bivalent: number analyzed (Participants) | 556 | 1103
  Month 25b: Bivalent | 1.8 | 0.0907
  Month 25b: Trivalent: number analyzed (Participants) | 556 | 1103
  Month 25b: Trivalent | 1.6 | 0.4
  Month 25b: Tetravalent: number analyzed (Participants) | 556 | 1102
  Month 25b: Tetravalent | 74.5 | 99.5
  Month 25b: At Least Bivalent: number analyzed (Participants) | 556 | 1103
  Month 25b: At Least Bivalent | 77.9 | 99.909
  Month 25b: At Least Trivalent: number analyzed (Participants) | 556 | 1103
  Month 25b: At Least Trivalent | 76.1 | 99.8

44. Other Pre Specified Outcome: Geometric Mean Titers (GMTs) of Neutralizing Antibodies for Each of the Four Dengue Serotypes During Parts 4 And 5
Description: GMTs of neutralizing antibodies were measured via MNT50. The four DENV serotypes are DENV-1, DENV-2, DENV-3 and DENV-4.
Time Frame: as for outcome 42
Population: as for outcome 43
Measure: Geometric Mean (95% Confidence Interval); unit: titres
Arm/Group | Placebo | TDV 0.5 mL
Number analyzed (Participants) | 597 | 1186
titres
  Day 1b: DENV-1 | 172.7 [137.8 to 216.5] | 374.7 [332.7 to 422.1]
  Day 1b: DENV-2 | 164.5 [133.2 to 203.2] | 609.4 [558.6 to 664.7]
  Day 1b: DENV-3 | 129.4 [105.0 to 159.4] | 305.2 [274.6 to 339.3]
  Day 1b: DENV-4 | 81.5 [67.8 to 98.1] | 172.9 [156.1 to 191.4]
  Month 1b: DENV-1: number analyzed (Participants) | 542 | 1075
  Month 1b: DENV-1 | 179.8 [142.4 to 227.0] | 1493.8 [1383.2 to 1613.3]
  Month 1b: DENV-2: number analyzed (Participants) | 542 | 1075
  Month 1b: DENV-2 | 174.8 [140.5 to 217.6] | 1611.5 [1492.1 to 1740.4]
  Month 1b: DENV-3: number analyzed (Participants) | 542 | 1075
  Month 1b: DENV-3 | 159.9 [128.4 to 199.0] | 1546.6 [1450.0 to 1649.6]
  Month 1b: DENV-4: number analyzed (Participants) | 542 | 1075
  Month 1b: DENV-4 | 87.3 [72.0 to 105.9] | 793.8 [742.5 to 848.7]
  Month 6b: DENV-1: number analyzed (Participants) | 562 | 1127
  Month 6b: DENV-1 | 191.5 [152.2 to 241.0] | 1000.9 [916.8 to 1092.7]
  Month 6b: DENV-2: number analyzed (Participants) | 562 | 1127
  Month 6b: DENV-2 | 208.0 [167.6 to 258.0] | 1167.2 [1080.8 to 1260.5]
  Month 6b: DENV-3: number analyzed (Participants) | 562 | 1127
  Month 6b: DENV-3 | 156.0 [126.1 to 192.9] | 851.0 [788.9 to 917.9]
  Month 6b: DENV-4: number analyzed (Participants) | 562 | 1127
  Month 6b: DENV-4 | 86.4 [71.9 to 103.9] | 457.6 [427.4 to 490.0]
  Month 13b: DENV-1: number analyzed (Participants) | 561 | 1122
  Month 13b: DENV-1 | 259.3 [204.8 to 328.4] | 949.1 [862.2 to 1044.7]
  Month 13b: DENV-2: number analyzed (Participants) | 561 | 1122
  Month 13b: DENV-2 | 248.9 [199.4 to 310.6] | 1003.2 [920.1 to 1093.9]
  Month 13b: DENV-3: number analyzed (Participants) | 561 | 1122
  Month 13b: DENV-3 | 199.1 [159.9 to 248.0] | 804.1 [739.2 to 874.8]
  Month 13b: DENV-4: number analyzed (Participants) | 561 | 1122
  Month 13b: DENV-4 | 115.0 [94.4 to 140.0] | 433.1 [401.2 to 467.6]
  Month 25b: DENV-1: number analyzed (Participants) | 556 | 1103
  Month 25b: DENV-1 | 293.8 [233.1 to 370.3] | 865.6 [782.7 to 957.2]
  Month 25b: DENV-2: number analyzed (Participants) | 556 | 1103
  Month 25b: DENV-2 | 278.5 [224.3 to 345.8] | 951.6 [873.0 to 1037.2]
  Month 25b: DENV-3: number analyzed (Participants) | 556 | 1102
  Month 25b: DENV-3 | 229.7 [185.5 to 284.3] | 688.3 [632.2 to 749.3]
  Month 25b: DENV-4: number analyzed (Participants) | 556 | 1103
  Month 25b: DENV-4 | 129.2 [106.8 to 156.3] | 387.9 [358.6 to 419.6]

45. Other Pre Specified Outcome: Geometric Mean Ratio (GMR) of Neutralizing Antibodies for Each Dengue Serotype
Description: The GMR is the geometric mean of the ratio of the two visits being compared.
Time Frame: Pre-booster Vaccination on Day 1b (Month 0b) versus post-booster vaccination on Day 30b (Month 1b) in Part 4
Population: PPSI-B: all participants in FASI-B who had no major protocol violations. FASI-B: all participants from FAS-B who were included in booster immunogenicity subset & for whom there is valid pre-booster measurement & at least 1 valid post-booster measurement for immunogenicity assessments. Overall number of participants analyzed: number of participants with data available for analyses. Number analyzed: number of participants with data available for analyses for specified category.
Measure: Geometric Mean (95% Confidence Interval); unit: unitless ratio
Arm/Group | Placebo | TDV 0.5 mL
Number analyzed (Participants) | 396 | 1067
unitless ratio
  DENV-1: number analyzed (Participants) | 383 | 1016
  DENV-1 | 0.9 [0.8 to 1.0] | 3.1 [2.8 to 3.4]
  DENV-2 | 0.9 [0.9 to 1.0] | 2.4 [2.3 to 2.6]
  DENV-3: number analyzed (Participants) | 375 | 1042
  DENV-3 | 1.1 [1.0 to 1.2] | 4.3 [3.9 to 4.7]
  DENV-4: number analyzed (Participants) | 365 | 1008
  DENV-4 | 0.9 [0.9 to 1.0] | 3.5 [3.2 to 3.9]

46. Other Pre Specified Outcome: GMR of Neutralizing Antibodies for Each Dengue Serotype
Description: The GMR is the geometric mean of the ratio of the two visits being compared.
Time Frame: Pre-booster Vaccination on Day 1b (Month 0b) versus post-booster vaccination on Day 180b (Month 6b) in Part 4
Population: as for outcome 45
Measure: Geometric Mean (95% Confidence Interval); unit: unitless ratio
Arm/Group | Placebo | TDV 0.5 mL
Number analyzed (Participants) | 408 | 1120
unitless ratio
  DENV-1: number analyzed (Participants) | 396 | 1064
  DENV-1 | 1.0 [0.9 to 1.1] | 2.2 [2.0 to 2.4]
  DENV-2 | 1.1 [1.0 to 1.3] | 1.8 [1.7 to 2.0]
  DENV-3: number analyzed (Participants) | 389 | 1094
  DENV-3 | 1.0 [0.9 to 1.1] | 2.5 [2.3 to 2.7]
  DENV-4: number analyzed (Participants) | 377 | 1052
  DENV-4 | 0.9 [0.8 to 1.0] | 2.1 [2.0 to 2.3]

47. Other Pre Specified Outcome: GMR of Neutralizing Antibodies for Each Dengue Serotype
Description: The geometric mean ratio is the geometric mean of the ratio of the two visits being compared.
Time Frame: Pre-booster Vaccination on Day 1b (Month 0b) versus post-booster vaccination on Day 395b (Month 13b) in Part 4
Population: as for outcome 45
Measure: Geometric Mean (95% Confidence Interval); unit: unitless ratio
Arm/Group | Placebo | TDV 0.5 mL
Number analyzed (Participants) | 408 | 1114
unitless ratio
  DENV-1: number analyzed (Participants) | 395 | 1060
  DENV-1 | 1.3 [1.1 to 1.5] | 2.1 [1.9 to 2.3]
  DENV-2 | 1.3 [1.1 to 1.5] | 1.6 [1.5 to 1.7]
  DENV-3: number analyzed (Participants) | 389 | 1088
  DENV-3 | 1.3 [1.1 to 1.5] | 2.4 [2.2 to 2.6]
  DENV-4: number analyzed (Participants) | 376 | 1047
  DENV-4 | 1.3 [1.1 to 1.4] | 2.0 [1.9 to 2.2]

48. Other Pre Specified Outcome: GMR of Neutralizing Antibodies for Each Dengue Serotype
Description: The geometric mean ratio is the geometric mean of the ratio of the two visits being compared.
Time Frame: Pre-booster Vaccination on Day 1b (Month 0b) versus post-booster vaccination on Day 720b (Month 25b) in Part 5
Population: as for outcome 45
Measure: Geometric Mean (95% Confidence Interval); unit: unitless ratio
Arm/Group | Placebo | TDV 0.5 mL
Number analyzed (Participants) | 398 | 1095
unitless ratio
  DENV-1: number analyzed (Participants) | 384 | 1043
  DENV-1 | 1.3 [1.2 to 1.5] | 2.0 [1.9 to 2.2]
  DENV-2 | 1.3 [1.1 to 1.5] | 1.6 [1.5 to 1.7]
  DENV-3: number analyzed (Participants) | 379 | 1068
  DENV-3 | 1.4 [1.2 to 1.6] | 2.1 [1.9 to 2.3]
  DENV-4: number analyzed (Participants) | 367 | 1028
  DENV-4 | 1.3 [1.1 to 1.5] | 1.9 [1.8 to 2.1]

ADVERSE EVENTS:
Time Frame: Part 1+ Part 2 combined: Deaths and SAEs from Day1 until end of Part 2(approx.21 months); Other AEs up to 28 days post first/second vaccination- i.e. only Part1; Part3: Deaths and SAEs during Part3(approx.3 years); no Other AEs collected during Part 3; Part 4+ Part 5 combined: Deaths and SAEs from booster vaccination (Day 1b) until end of Part 5 [approx. 25 months]; Other AEs up to 28 days post booster vaccination- i.e. only Part 4).
Description: As pre-specified in protocol, AEs are reported separately for Placebo and TDV arms of each Part. For Part 1-3: Safety Set. For Part 4-5: Safety Set-Booster.
Groups:
- TDV (Part 1): Participants received TDV, 0.5 mL, SC injection on Day 1 (Month 0) and Day 90 (Month 3) in Part 1 of the study.
- Placebo (Part 2); TDV (Part 2): Participants went through extended follow-up period for six months up to Month 21 in Part 2 of the study.
- Placebo (Part 3): Participants went through long-term follow-up (3 years) to evaluate the safety.
- TDV (Part 3): Participants eligible for Booster Phase received placebo matching TDV, SC injection, based on the randomization on Day 1 (Month 0) in Part 4 of the study.
- Placebo (Part 4): Participants eligible for Booster Phase received placebo matching TDV, SC injection, based on the randomization on Day 1 (Month 0)in Part 4 of the study.
- TDV (Part 4): Participants eligible for Booster Phase received TDV, SC injection, based on the randomization on Day 1 (Month 0) in Part 4 of the study.
- Placebo (Part 5); TDV (Part 5): Participants went through extended follow-up period for 1 year up to Month 25b in Part 5 of the study.
Arm/Group | Placebo | TDV (Part 1) | Placebo (Part 2) | TDV (Part 2) | Placebo (Part 3) | TDV (Part 3) | Placebo (Part 4) | TDV (Part 4) | Placebo (Part 5) | TDV (Part 5)
All-Cause Mortality (participants affected / at risk) | 8/6687 | 22/13380 | 7/6519 | 18/13033 | 7/6487 | 17/12961 | 1/2985 | 6/5990 | 0/2939 | 3/5889
Serious Adverse Events (participants affected / at risk) | 256/6687 | 414/13380 | 82/6519 | 152/13033 | 397/6487 | 666/12961 | 126/2985 | 161/5990 | 73/2939 | 109/5889
Other Adverse Events (participants affected / at risk) | 527/6687 | 1260/13380 | 0/6519 | 0/13033 | 0/6487 | 0/12961 | 149/2985 | 409/5990 | 0/2939 | 0/5889
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=6687) | TDV (Part 1) (N=13380) | Placebo (Part 2) (N=6519) | TDV (Part 2) (N=13033) | Placebo (Part 3) (N=6487) | TDV (Part 3) (N=12961) | Placebo (Part 4) (N=2985) | TDV (Part 4) (N=5990) | Placebo (Part 5) (N=2939) | TDV (Part 5) (N=5889)
Abdominal abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 4 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 3 | 1 | 1 | 3 | 4 | 2 | 1 | 1 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abnormal uterine bleeding (Reproductive system and breast disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abnormal weight gain (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abortion (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abortion complete (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Abortion incomplete (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Abortion induced (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abortion infected (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 2 | 1 | 2 | 7 | 6 | 0 | 1 | 3 | 0
Abortion spontaneous incomplete (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Abortion threatened (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Abscess jaw (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abscess limb (Infections and infestations) | 2 | 5 | 0 | 1 | 2 | 7 | 0 | 0 | 0 | 2
Abscess neck (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Abscess of external ear (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abscess soft tissue (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acarodermatitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Accident at work (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Accidental exposure to product by child (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acid peptic disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Acute disseminated encephalomyelitis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute psychosis (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute sinusitis (Infections and infestations) | 1 | 0 | 2 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Adjustment disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Adjustment disorder with depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Aggression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Allergy to arthropod bite (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Alveolar rhabdomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Amaurosis (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Amniotic cavity infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Amoebiasis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Amoebic dysentery (Infections and infestations) | 2 | 1 | 0 | 1 | 1 | 6 | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Anaemia of pregnancy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 2 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Anaphylactic shock (Immune system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Anembryonic gestation (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Animal bite (Injury, poisoning and procedural complications) | 4 | 8 | 1 | 2 | 3 | 10 | 0 | 2 | 2 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Antisocial behaviour (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0
Anxiety disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aortic valve incompetence (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Appendiceal abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 14 | 30 | 6 | 14 | 27 | 60 | 5 | 7 | 4 | 12
Appendicitis perforated (Infections and infestations) | 0 | 2 | 0 | 3 | 6 | 7 | 0 | 3 | 0 | 2
Aqueductal stenosis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arboviral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arteriovenous malformation (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthritis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ascariasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 7 | 1 | 7 | 2 | 5 | 0 | 3 | 0 | 2
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1 | 2 | 2 | 0 | 1 | 0 | 1 | 1
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Atrial septal defect (Congenital, familial and genetic disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atypical pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Avulsion fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Back injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bacterial infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bacterial sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bacterial vaginosis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bacteriuria (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Balanoposthitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bartholin's abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Behaviour disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Behcet's syndrome (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bell's palsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Benign hydatidiform mole (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bipolar I disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blindness traumatic (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood loss anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Brain hypoxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Breast abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0
Breast cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 4 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 0
Bronchitis viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bullous impetigo (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Burkholderia pseudomallei infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Burn infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Burns second degree (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 24 | 69 | 39 | 65 | 0 | 1
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 3 | 7 | 0 | 1 | 0 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Carcinoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 10 | 1 | 3 | 7 | 15 | 2 | 3 | 1 | 0
Cellulitis orbital (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cephalo-pelvic disproportion (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cerebellar infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cerebral arteriovenous malformation haemorrhagic (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cerebral venous thrombosis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cerebrovascular arteriovenous malformation (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chemical burn of oral cavity (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chest injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chikungunya virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Cholangitis sclerosing (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Cholera (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Completed suicide (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 4 | 0 | 0 | 0 | 0
Complicated appendicitis (Infections and infestations) | 1 | 6 | 1 | 2 | 7 | 12 | 4 | 2 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 3 | 0 | 1 | 2 | 1 | 0 | 0 | 2 | 0
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Conjunctivitis allergic (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 1 | 1 | 2 | 3 | 5 | 1 | 1 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Corneal opacity (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Coronavirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 3 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 1
Craniofacial fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0
Croup infectious (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cryptorchism (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cushing's syndrome (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cutaneous T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 3 | 3 | 0 | 0 | 0 | 0
Dengue fever (Infections and infestations) | 52 | 13 | 10 | 9 | 83 | 56 | 32 | 7 | 17 | 9
Dengue haemorrhagic fever (Infections and infestations) | 19 | 4 | 6 | 1 | 12 | 9 | 4 | 0 | 3 | 0
Depression (Psychiatric disorders) | 0 | 2 | 0 | 1 | 2 | 7 | 2 | 1 | 0 | 0
Dermatitis infected (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dermoid cyst (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Desmoplastic small round cell tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Device extrusion (Product Issues) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Device malfunction (Product Issues) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 2 | 0 | 1 | 1 | 3 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Diplegia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Disruptive mood dysregulation disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Disseminated tuberculosis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Drowning (General disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1
Drug abuse (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysentery (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Electric injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electric shock (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Electrical burn (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
End stage renal disease (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Enteritis infectious (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0
Ependymoma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epididymitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Epidural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1
Epiphyseal injury (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Epiphysiolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Erythema annulare (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Erythema infectiosum (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 3 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Exostosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Exposure to communicable disease (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Extradural abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Extradural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Extremity contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Extremity necrosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eye infection gonococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eye injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eyelid injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Face injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 1 | 1 | 0 | 4 | 3 | 1 | 1 | 0
False labour (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
False positive investigation result (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Familial periodic paralysis (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Febrile convulsion (Nervous system disorders) | 1 | 4 | 1 | 2 | 1 | 1 | 1 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 3 | 0 | 0 | 2 | 3 | 0 | 0 | 0 | 0
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Focal peritonitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Food allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 3 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 3 | 0 | 0 | 1 | 2 | 2
Forearm fracture (Injury, poisoning and procedural complications) | 2 | 8 | 1 | 2 | 2 | 9 | 4 | 3 | 2 | 1
Foreign body in gastrointestinal tract (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fractured coccyx (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gangrene (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 6 | 3 | 2 | 3 | 6 | 0 | 0 | 0 | 1
Gastritis erosive (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 8 | 29 | 2 | 7 | 11 | 18 | 2 | 1 | 0 | 4
Gastroenteritis bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Gastroenteritis salmonella (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis shigella (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 3 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Gastrointestinal bacterial infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Giardiasis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Glomerulonephritis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Glomerulonephritis acute (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0
Glomerulonephritis chronic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Glomerulonephritis proliferative (Renal and urinary disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Glomerulonephritis rapidly progressive (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Goitre (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Greater trochanteric pain syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Groin abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Guillain-Barre syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Gun shot wound (Injury, poisoning and procedural complications) | 0 | 3 | 1 | 0 | 3 | 3 | 0 | 0 | 0 | 1
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 2 | 2 | 0 | 3 | 5 | 1 | 0 | 1 | 1
Hand-foot-and-mouth disease (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hanging (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 3 | 4 | 0 | 0 | 0 | 3 | 1 | 1 | 0 | 1
Headache (Nervous system disorders) | 0 | 3 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Hepatic rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatitis A (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0
Hepatitis acute (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatitis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0
Hepatosplenomegaly (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Herpes simplex encephalitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
High risk pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
High risk sexual behaviour (Social circumstances) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 3 | 10 | 0 | 0 | 2 | 7 | 1 | 0 | 1 | 0
Hydrocephalus (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperemesis gravidarum (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 2 | 2 | 0 | 0 | 0 | 0
Hypertensive nephropathy (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertensive urgency (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Idiopathic generalised epilepsy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
IgA nephropathy (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ileus paralytic (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ilium fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Immune thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Impetigo (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Incarcerated umbilical hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infected bite (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Infectious mononucleosis (Infections and infestations) | 0 | 3 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Infective exacerbation of asthma (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infective myositis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Inflammatory myofibroblastic tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 7 | 14 | 5 | 6 | 9 | 12 | 1 | 0 | 1 | 3
Influenza like illness (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 1 | 2 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Intentional self-injury (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 1
Intra-abdominal fluid collection (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Joint abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Juvenile idiopathic arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Kawasaki's disease (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Knee deformity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Labour complication (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leptospirosis (Infections and infestations) | 2 | 2 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lichen planus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Ligament injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Limb crushing injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 3 | 2 | 4 | 0 | 0 | 0 | 1
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0
Lip injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Liver contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Localised infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 4 | 0 | 1 | 1 | 1
Lower respiratory tract infection (Infections and infestations) | 3 | 10 | 1 | 3 | 3 | 3 | 0 | 1 | 1 | 0
Ludwig angina (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lung abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lupus nephritis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Lupus pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lymph gland infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lymph node tuberculosis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 2 | 2 | 1 | 0 | 1 | 0 | 0
Lymphadenitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lymphoid hyperplasia of intestine (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Major depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 1
Malaria (Infections and infestations) | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mania (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mastoiditis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Measles (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mechanical ileus (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Medulloblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Meningitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Meningitis aseptic (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Meningitis tuberculous (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mesenteric cyst (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mesenteric lymphadenitis (Blood and lymphatic system disorders) | 0 | 5 | 0 | 2 | 0 | 4 | 0 | 0 | 2 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Metabolic dysfunction-associated steatohepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Metabolic syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 3 | 0 | 1 | 0 | 0
Mixed anxiety and depressive disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 3 | 1 | 0 | 0 | 4 | 1 | 0 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscle abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscle injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscular dystrophy (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Myelopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 3 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Neck injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nephritic syndrome (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Nephrotic syndrome (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Obstetric infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Obstructive sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Open globe injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Oppositional defiant disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Optic neuritis (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Orbital myositis (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Orchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Organ failure (General disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Osteochondroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Osteomyelitis chronic (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Otitis media acute (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ovarian germ cell endodermal sinus tumour stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Ovulation pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pancreatic injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pancreatic pseudocyst (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paranasal sinus abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Parasite allergy (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Parasitic gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0
Parotitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Partial seizures (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pelvic abscess (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pelvic inflammatory disease (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 2
Penetrating abdominal trauma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Penile adhesion (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Peptic ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Perineal injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Periorbital abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Periorbital cellulitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0
Peritonsillar abscess (Infections and infestations) | 0 | 3 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 3 | 3 | 2 | 0 | 1 | 0 | 0
Pharyngitis bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pharyngotonsillitis (Infections and infestations) | 2 | 3 | 0 | 2 | 1 | 2 | 0 | 0 | 1 | 0
Phimosis (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Physical assault (Social circumstances) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pilonidal disease (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Placental insufficiency (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 8 | 10 | 7 | 6 | 8 | 20 | 0 | 2 | 0 | 3
Pneumonia bacterial (Infections and infestations) | 2 | 2 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0
Pneumonia influenzal (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia mycoplasmal (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Polyarteritis nodosa (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Polyhydramnios (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Portal hypertension (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Post infection glomerulonephritis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Post procedural discharge (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post procedural infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Post streptococcal glomerulonephritis (Renal and urinary disorders) | 0 | 5 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Post-traumatic headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Postoperative adhesion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0 | 1 | 0 | 2 | 4 | 0 | 0 | 0 | 0
Postpartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 1
Postpartum sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 1 | 4 | 9 | 0 | 0 | 0 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Premature delivery (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 3 | 8 | 0 | 1 | 2 | 0
Premature labour (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 3 | 2 | 0 | 0 | 0 | 0
Premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 1 | 1
Premature separation of placenta (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Preterm premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pseudomembranous colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Psychiatric symptom (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Psychogenic seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Puerperal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 4 | 0 | 1 | 0 | 1
Pustule (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyelocaliectasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 1 | 0 | 0 | 4 | 2 | 2 | 0 | 0 | 0
Pyoderma (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 5 | 0 | 2 | 1 | 1 | 1 | 0 | 1 | 0
Quadriparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 7 | 3 | 1 | 1 | 2 | 12 | 1 | 3 | 0 | 2
Rectal polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Red blood cell sedimentation rate increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Refraction disorder (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Retinal haemorrhage (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rheumatic fever (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rheumatic heart disease (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rickettsiosis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 8 | 1 | 1 | 2 | 9 | 3 | 3 | 3 | 6
Ruptured cerebral aneurysm (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ruptured ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
SARS-CoV-2 sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Salpingitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Scarlet fever (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Schwannoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Scrotal pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 1 | 2 | 0 | 1 | 1 | 3 | 0 | 0 | 0 | 0
Self-destructive behaviour (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1 | 1 | 4 | 0 | 0 | 1 | 0 | 0
Septic phlebitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Septic shock (Infections and infestations) | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Serositis (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Serotonin syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sexual abuse (Social circumstances) | 3 | 1 | 0 | 4 | 0 | 1 | 0 | 1 | 0 | 1
Shock (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Shunt malfunction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Simple partial seizures (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sinus node dysfunction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sinus polyp (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Sinusitis bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin injury (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 2 | 3 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Skull fracture (Injury, poisoning and procedural complications) | 0 | 3 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Skull fractured base (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Small intestinal perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Snake bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Spinal cord injury thoracic (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Splenic rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Spondylitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sports injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Stab wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Staphylococcal abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Status migrainosus (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 2 | 0 | 1 | 0 | 4 | 0 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Subgaleal haematoma (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Substance use (Social circumstances) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Substance use disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Suicidal behaviour (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Suicide attempt (Psychiatric disorders) | 1 | 2 | 0 | 2 | 5 | 5 | 0 | 1 | 2 | 1
Superinfection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Suspected COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 2 | 2 | 0 | 0 | 2 | 3 | 0 | 2 | 0 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syphilis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Systemic viral infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tendon injury (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tension headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Testicular injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Testicular torsion (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 1 | 3 | 1 | 0 | 1 | 0
Thalassaemia alpha (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Threatened labour (Pregnancy, puerperium and perinatal conditions) | 0 | 2 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 2 | 2 | 1 | 0 | 2 | 5 | 0 | 4 | 0 | 0
Tinea capitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 1 | 3 | 1 | 2 | 3 | 2 | 0 | 0 | 0 | 1
Tonsillitis bacterial (Infections and infestations) | 2 | 4 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 2 | 5 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 2 | 1
Traumatic delivery (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Traumatic haemothorax (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Traumatic liver injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Traumatic lung injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Type I hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Typhoid fever (Infections and infestations) | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ulcerated haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Umbilical cord prolapse (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0
Unstable foetal lie (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 5 | 3 | 1 | 0 | 4 | 9 | 0 | 0 | 1 | 2
Upper respiratory tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urethral caruncle (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urethritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary bladder rupture (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 5 | 9 | 2 | 4 | 15 | 20 | 0 | 3 | 2 | 3
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 4 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1
Vaginal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Varicella (Infections and infestations) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vasculitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Venom poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ventricular arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Victim of crime (Social circumstances) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Victim of sexual abuse (Social circumstances) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Viral infection (Infections and infestations) | 19 | 23 | 4 | 3 | 17 | 16 | 3 | 1 | 5 | 3
Viral myocarditis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Viral pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Viral rash (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Vulval haematoma (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vulvovaginal injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 3 | 1 | 1 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=6687) | TDV (Part 1) (N=13380) | Placebo (Part 2) (N=6519) | TDV (Part 2) (N=13033) | Placebo (Part 3) (N=6487) | TDV (Part 3) (N=12961) | Placebo (Part 4) (N=2985) | TDV (Part 4) (N=5990) | Placebo (Part 5) (N=2939) | TDV (Part 5) (N=5889)
Headache (Nervous system disorders) | 337 | 736 | 0 | 0 | 0 | 0 | 82 | 206 | 0 | 0
Pain (General disorders) | 363 | 1011 | 0 | 0 | 0 | 0 | 113 | 340 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.

DOCUMENTS (2):
  • Study Protocol (2021-09-14): https://cdn.clinicaltrials.gov/large-docs/27/NCT02747927/Prot_004.pdf
  • Statistical Analysis Plan (2020-09-24): https://cdn.clinicaltrials.gov/large-docs/27/NCT02747927/SAP_003.pdf